#### GTI1401

A Multi-Center, Open-Label, Phase I/II Study to Evaluate the Safety and Pharmacokinetics of Weekly Intravenous Infusions of Alpha-1 MP in Japanese Subjects with a<sub>1</sub>-Antitrypsin Deficiency

Protocol Version: GTI1401 Version 1.5J (05July2016)

#### GTI1401-OLE

A Multi-Center, Open-Label Study to Evaluate the Long-term Safety of Weekly Intravenous Infusions of Alpha-1 MP in Japanese Subjects with a1-Antitrypsin Deficiency

Protocol Version: GTI1401-OLE Version 1.3J (07July2016)

Statistical Analysis Plan

Version 1.0 / 21MAR2017 Prepared by:

Grifols Therapeutics Inc.

79 TW Alexander Drive Research Triangle Park, NC 27709

Issued by:

Date: Mar, 23,2017

Upon review of this document, including table, listing, and figure shells, the undersigned approves the statistical analysis plan. The analysis methods and data presentation are acceptable, and the table, listing, and figure production can begin.

Approved by:

Approved by:

PhD Pharm.D.

Date: Mar 21 2017

Date: Man 21 2017

Grifols Inc. GT11401/GT11401-OLE

Approved by:

Approved by:

Ph.D.

Statistical Analysis Plan 21MAR2017

Date: 144/12/2017

Date: Mar/ 23/ 2017

Date: 3 /23/2017

# TABLE OF CONTENTS

| 1 | | PURPOSE OF THE ANALYSIS | 7 |
|---|---|---|---|
| 2 | | INTRODUCTION | 7 |
| 3 | | OBJECTIVES | 8 |
| | 3.1<br>3.2<br>3.3 | PRIMARY OBJECTIVES | 8 |
| 4 | | INVESTIGATIONAL PLAN | 9 |
| | 4.1<br>4.2 | STUDY DESIGN AND PLAN STUDY VARIABLES | |
| 5 | | GENERAL STATISTICAL CONSIDERATIONS | 13 |
| | 5.2<br>5.3<br>5.4<br>5.5<br>5.6 | PK Data Handling Handling of Missing values Safety Data Handling Sample Size Rounding Analysis Populations Denominator | 13<br>13<br>14<br>14<br>15 |
| 6 | | SUBJECT DISPOSITION | 16 |
| 7 | | PROTOCOL DEVIATIONS | 16 |
| 8 | | DEMOGRAPHICS | 17 |
| 9 | | TREATMENTS AND MEDICATIONS | 18 |
| | 9.1<br>9.2<br>9.3 | PRIOR AND CONCOMITANT MEDICATIONS EXTENT OF EXPOSURE TREATMENT COMPLIANCE | 18<br>20 |
| 1( | ) | EXPLORATORY ANALYSIS | |
| | 10.1<br>10.2 | PK ANALYSIS (GTI1401 ONLY) | |
| 11 | | SAFETY ANALYSIS | 27 |
| | | ADVERSE EVENTS LABORATORY TESTS VITAL SIGNS ELECTROCARDIOGRAM URINE COTININE TEST | 30<br>32<br>33<br>33 |
| | 11.6 | PULMONARY FUNCTION TESTS | 34 |

## Statistical Analysis Plan 21MAR2017

| 11.7 | Pregnancy Tests | . 34 |
|------|-----------------------------|------|
| 11.8 | CT Scan | 35 |
| | PHYSICAL EXAMINATION | |
| 12 | INTERIM ANALYSIS | 35 |
| 13 | CHANGES IN PLANNED ANALYSIS | 35 |

#### LIST OF ABBREVIATIONS

AATD Alpha<sub>1</sub>-antitrypsin deficiency

ADR Adverse drug reaction

AE Adverse event

Alpha-1 MP Alpha<sub>1</sub>-proteinase inhibitor (human), modified process

Alpha<sub>1</sub>-PI Alpha<sub>1</sub>-proteinase inhibitor

ALT Alanine aminotransferase

AST Aspartate transaminase

ATS American Thoracic Society

AUC Area under the concentration-time curve

BLQ Below limit of quantification

C<sub>max</sub> Maximum concentration

COPD Chronic obstructive pulmonary disease

CRF Case report form

CV Coefficient of variation

FEV<sub>1</sub> Forced expiratory volume in 1 second

FVC Forced vital capacity

GCP Good Clinical Practice

HAV Hepatitis A virus
HBV Hepatitis B virus
HCV Hepatitis C virus

HIV Human immunodeficiency virus

IgA Immunoglobulin A
IgG Immunoglobulin G
IgM Immunoglobulin M

MedDRA® Medical Dictionary for Regulatory Activities

NE Neutrophil elastase

PFT Pulmonary Function Test

PI\*MM Proteinase inhibitor homozygote for normal M allele

PI\*(null)(null) Proteinase inhibitor homozygote for (null) allele

PI\*SZ Proteinase inhibitor heterozygote for S and Z deficiency alleles

PI\*Z Proteinase inhibitor Z deficiency allele

PI\*ZZ Proteinase inhibitor homozygote for Z deficiency allele

pH Potential of hydrogen; acidity/alkalinity measure

PK Pharmacokinetics

SAE Serious adverse event
SAP Statistical analysis plan

SD Standard deviation t½ Terminal half-life

TEAE Treatment-emergent adverse event

tmax Time to reach Cmax

US United States

WHO-DD World health organization drug dictionary

## 1 Purpose of the Analysis

The purpose of this statistical analysis plan (SAP) is to outline the planned analyses to support the completion of the clinical study report (CSR) for protocol GTI1401 and GTI1401-OLE. The planned analyses identified in this SAP will be included in regulatory submissions and/or future manuscripts. Exploratory analyses not identified or defined in this SAP may be performed to support the clinical development program. Any post hoc or unplanned analyses performed and not identified in this SAP will be documented in the respective CSR.

#### 2 Introduction

Alpha<sub>1</sub>-antitrypsin deficiency (AATD) is a genetic disorder in which mutations of the SERPINA1 gene (a member of the SERPIN, serine protease inhibitor gene family) lead to a reduced serum level of the serine protease inhibitor called alpha<sub>1</sub>-proteinase inhibitor (alpha<sub>1</sub>-PI) or, historically, alpha<sub>1</sub>-antitrypsin. AATD manifests clinically as pulmonary emphysema, chronic obstructive pulmonary disease (COPD), and liver cirrhosis.

The most frequent mutation causing severe AATD is called PI\*Z and was first described in a Swedish patient with emphysema. PI\*MM (normal) individuals have serum alpha<sub>1</sub>-PI levels in the range of 20 to 53  $\mu$ M; however, PI\*ZZ (homozygous abnormal) individuals with AATD have serum alpha<sub>1</sub>-PI levels in the range of 2 to 10.2  $\mu$ M. The estimated world-wide prevalence of PI\*ZZ and PI\*SZ (heterozygous abnormal) individuals is approximately 163,700 and 903,000, respectively.

Like other hereditary disorders, AATD is relatively rare (e.g., has orphan drug designation); however, it is extremely rare among Asians. In 2000, a survey supported by the Japanese Ministry of Health and Welfare identified only 16 individuals in Japan with documented AATD. AATD in Japanese patients exhibits unique features compared to AATD in Caucasians, including the lack of a PI\*Z variant and a high incidence of the S<sub>iiyama</sub> deficiency AATD variant. In Japanese patients homozygous for the S<sub>iiyama</sub> variant, serum alpha<sub>1</sub>-PI levels are in the range of 2.1 to 7.7 μM. Japanese normal individuals have serum alpha<sub>1</sub>-PI levels in the range of 21 to 34 μM (94 to 150 mg/dL as measured by nephelometry, which is used as the laboratory test standard values).

Augmentation therapy with intravenous (IV) alpha<sub>1</sub>-PI is administered in patients with AATD to increase the low serum concentrations in this patient population. This usage is intended to bolster the protective protease inhibitory shield against increased numbers of lung neutrophils releasing increased concentrations of NE, leading to a corrected protease: antiprotease imbalance. The restored antiprotease shield then protects the lung from elastolytic damage and slows the development of pulmonary emphysema.

Alpha<sub>1</sub>-PI (human), Prolastin<sup>®</sup>, was licensed for use as augmentation therapy for AATD, at a dose of 60 mg/kg weekly, in the United States (US) in 1987 and in Germany in 1988. To date, Prolastin<sup>®</sup> has been approved in 20 countries including the United States and

European countries. Subsequently, Grifols incorporated modifications into the Prolastin manufacturing process to produce alpha<sub>1</sub>-PI (human), modified process (Alpha-1 MP). This modified process results in an increased yield of alpha<sub>1</sub>-PI and a product with twice the alpha<sub>1</sub>-PI concentration with an improved pathogen safety profile and higher purity compared to Prolastin. Alpha-1 MP is approved for 60 mg/kg weekly IV administration in the US, Canada, Argentina, Columbia, Turkey, Chile and Australia for the treatment of patients with severe AATD and clinically evident emphysema under the trade name Prolastin®-C.

Japanese patients with AATD exhibit very different genotypes of AATD compared to the rest of the world, and the number of Japanese patients with AATD is extremely small. These subjects can exhibit symptoms of emphysema-typed COPD and therefore, will have clinically evident emphysema and along with alpha<sub>1</sub>-PI deficiency. The safety and PK of augmentation therapy with Alpha-1 MP to increase serum alpha<sub>1</sub>-PI levels has not been evaluated in Japanese patients with AATD. Thus, Grifols Therapeutics Inc. and Grifols Japan K.K. is conducting a study to assess the safety and PK of 60 mg/kg Alpha-1 MP administered by weekly IV infusions over 8 weeks in Japanese subjects with AATD.

## 3 Objectives

## 3.1 Primary Objectives

The primary objective of GTI1401 study is to evaluate the safety of 60 mg/kg Alpha-1 MP administered by weekly IV infusions over eight weeks in Japanese subjects with AATD.

The primary objective of GTI1401-OLE study is to evaluate the long-term safety of 60 mg/kg Alpha-1 MP administered by weekly IV infusions for approximately one year or longer (can be renewed annually with the consent of the subjects) in adult subjects with AATD in Japan.

## 3.2 Secondary Objectives

The secondary objective of GTI1401 study is to evaluate the trough level of total alpha<sub>1</sub>-PI for weekly IV infusions of 60 mg/kg Alpha-1 MP in Japanese subjects with AATD.

The secondary objective of GTI1401-OLE study is not set up.

## 3.3 Exploratory Objectives

The exploratory objective of GTI1401 is to measure the following PK parameters for Alpha<sub>1</sub>-PI at steady state at the end of the 8-week treatment period.

• AUC<sub>0-7 days</sub>

Area under the concentration-time curve (AUC) from Day 0 to Day 7, calculated at steady state at the end of the 8-week treatment period.

- C<sub>max</sub>
   Maximum concentration
- $t_{max}$ The observed time to reach  $C_{max}$
- t<sub>1/2</sub>
  Terminal half-life

The exploratory objective of GTI1401-OLE is to perform CT scan (densitometry) at Ext Week 52. The CT scan data will be accumulated for the future evaluation of lung density.

• CT scan (densitometry)

Note: Subjects will undergo CT scanning for diagnosis of clinically apparent pulmonary emphysema in GTI1401 study. This CT scan data will also serve as the baseline measurement of lung density for GTI1401-OLE study.

## 4 Investigational Plan

## 4.1 Study Design and Plan

GTI1401 study is a multi-center, open-label, trial to evaluate the safety and PK of weekly IV infusions of 60 mg/kg Alpha-1 MP in Japanese subjects with AATD. At least three adult subjects will be enrolled in the study. The study consists of an up to three-week Screening Period, and an eight-week open-label Treatment Period including a one-week PK Assessment Period after the last infusion. At the Week 9 visit when the PK evaluation period is completed, subjects will be asked whether they would like to participate in an extension trial (GTI1401-OLE). For subjects not intending to participate in the extension trial, the date of follow-up/study completion visit (30 days [4 weeks] after the last dose of the investigational drug) will be arranged. The total duration of study participation for subjects who complete the study will be up to 14 weeks.

After providing informed consent at the Screening Visit, subjects will be evaluated for study eligibility during the Screening Period (up to three weeks); for study inclusion and exclusion criteria. Eligible subjects will enter the eight-week Treatment Period to receive a total of eight weekly IV infusions of 60 mg/kg Alpha-1 MP; subjects will receive their first infusion of Alpha-1 MP at the Week 1 (Baseline) Visit. During the Treatment Period, weekly infusions of Alpha-1 MP will be performed at the study site during scheduled study visits at Weeks 1 (Baseline), 2, 3, 4, 5, 6, 7, and 8. Subjects will receive their last infusion of Alpha-1 MP at the Week 8 Visit and will then enter the one-week

PK Assessment Period. During the PK Assessment Period, subjects have a last PK blood sampling study visit at Week 9. A Follow-Up/Final Visit (30 days [4 weeks] post last study drug infusion) will occur for subjects who will not participate in Study GTI1401-OLE.

All subjects will have a blood sample collected at Weeks 1 (Baseline), 7, and 8 (prior to the infusion of Alpha-1 MP) and Week 9 which will be used for the measurement of trough alpha<sub>1</sub>-PI levels.

Blood samples for PK parameters will be collected beginning at Week 8 and the collection of blood samples will extend into Week 9. The pre-infusion serial PK sample at Week 8 and the last serial PK sample (7 days after the Week 8 infusion) at Week 9 will also serve as trough blood samples for Weeks 8 and 9. The specific timing of all 10 serial blood samples includes:

- Immediately prior to infusion
- Immediately after infusion completion (after sodium chloride [NaCl] flush) (0 hour)
- 15 minutes after infusion completion
- 2 hours after infusion completion
- 4 hours after infusion completion
- 8 hours after infusion completion
- 24±4 hours (1 day after infusion completion)
- 48±4 hours (2 days after infusion completion)
- 120 hours  $\pm$  1 day (5 days after infusion completion)
- 168 hours  $\pm$  1 day (7 days after infusion completion) (Week 9 Visit)

At the Week 9 visit, subjects have the option to participate in an open-label extension (OLE) study (GTI1401-OLE) in which subjects, if they opt to enroll, will continue to receive 60 mg/kg Alpha-1 MP for at least another year (with the optional subsequent annual extensions) to assess the long-term safety of Alpha-1 MP. Week 9 of the GTI1401 study is also the first week of the extension study (GTI1401-OLE). If subjects do not opt to participate in Study GTI140-OLE, they will come back to the clinic 30 days (4 weeks) after the last Alpha-1 MP infusion for the Follow-Up/End of Study Visit (Week 12).

A schematic of the overall study design is shown in Figure 1 below. The schedule of events for GTI1401 and GTI1401-OLE studies can be found in appendix 1 and appendix 2.



 <sup>&</sup>lt;sup>a</sup> Final Visit/Early Termination = Follow-up/Final Evaluation Visit. Subjects who discontinue early from the study will need to complete this study visit 30days (4 weeks) after the last study drug infusion.
 <sup>b</sup> At the Week 9 Visit, subjects will be given the option to participate in the GTI1401-OLE. If they are enrolled in Study GTI1401-OLE, the Week 9 visit will be their End of Study Visit of GTI1401 study.

Figure 1 Overall Study Schema

#### 4.2 Study Variables

No efficacy variables will be assessed for the studies. The variables to be assessed for GTI1401 and GTI1401-OLE studies are as follows:

- Adverse events, ADRs, serious AEs (SAEs), and discontinuations due to AEs or SAEs
- Vital signs (heart rate, blood pressure, respiratory rate, and temperature)
- COPD exacerbations
- Pulmonary function tests:
  - o Forced Expiratory Volume in 1 second (FEV<sub>1</sub>)
  - o Forced Vital Capacity (FVC)
- Clinical laboratory parameters:
  - Chemistry
  - Hematology
  - Urinalysis
- Alpha<sub>1</sub>-PI trough level
- PK parameters (GTI1401 study only):
  - o AUC<sub>0-7 days</sub>
  - o C<sub>max</sub>
  - $\circ$   $t_{max}$

Grifols Therapeutics Inc. Statistical Analysis Plan
GTI1401/ GTI1401-OLE 21MAR2017

 $\circ \quad t_{\frac{1}{2}}$ 

• CT scan (densitometry)

#### 5 General Statistical Considerations

All analyses will be conducted using SAS Version 9.3 or higher.

Pharmacokinetic evaluations, descriptive statistical analysis of concentrations and PK parameters according to non-compartmental standard methods, as well as graphical representation of concentrations will be performed using the computer program Pharsight Phoenix WinNonlin (Version 6.1 or higher).

Unless otherwise specified, the results from GTI1401 and GTI1401-OLE will be presented separately.

Unless otherwise noted, for continuous variables, descriptive statistics will include the number of non-missing values, mean, standard deviation, median, minimum and maximum. For categorical variables, descriptive statistics will include counts and percentages per category.

## 5.1 PK Data Handling

For PK parameter estimation, the actual sample time instead of nominal time will be used. For the last time point (168 hours post infusion), if the actual time deviates from the scheduled time, the interpolation or extrapolation will be used to obtain the AUC<sub>0-7days</sub>.

When BLQ values are recorded, adopt the half value of the readable numeric value (2.5 mg/dL) for summarizing data.

#### 5.2 Handling of Missing values

Missing values will not be imputed unless otherwise specified.

For Adverse Event

Any missing severity/relationship will be accounted as "worst case" as related in the tables.

#### 5.3 Safety Data Handling

#### 5.3.1 Definition of Baseline

Baseline evaluations will be those collected (non-missing) closest to and prior to the first study drug infusion, which will be conducted –within 21 days of Week 1. For both GTI1401 and GTI1401-OLE, the baseline is the baseline visit at Week 1 in GTI1401 study.

For Pulmonary Function Tests

Values collected at "PRE-BRONCHODILATOR" time-point in screening visit will be defined as baseline for "PRE-BRONCHODILATOR". Also values collected at "POST-BRONCHODILATOR" time-point in screening visit will be defined as baseline for "POST-BRONCHODILATOR".

#### 5.3.2 Visit Windows for Safety Analyses

The date of all visits after the screening visit and the Week 1 (baseline) visit will be arranged within a time window of  $\pm 1$  day.

If an observation is missing at a specific scheduled visit, the value at that visit will be set to missing.

Visit recorded on CRF will be used as Analysis visit except Baseline visit.

#### 5.3.3 Unscheduled Visit

Data collected as unscheduled visits will not be used for the tables but presented in the listing and subject data plot.

#### 5.3.4 Follow-Up/End of Study Visit

30 days [4 weeks] after the completion of the last Alpha-1 MP infusion (Week 8) and 3 weeks after the Week 9 Visit, those subjects who do not participate in Study GTI1401-OLE will go to the clinic to complete a Follow-Up/End of Study Visit (Week 12). The Week 12 Visit should be scheduled at the protocol-specified study week relative to the date of the Week 1 (Baseline) Visit  $\pm$  1 day. The data collected during Follow-Up/End of Study Visit (Week 12) are included in Table and Listing for Safety Analysis and Concomitant Medication.

#### 5.4 Sample Size

The targeted sample size is at least 3 subjects. Sample size was chosen based on clinical considerations and the number of available Japanese patients with AATD, not on a formal sample size calculation.

#### 5.5 Rounding

In listings, data will be presented with the same precision as the original data; at the output creation stage, derived data will be rounded for presentation purposes.

For all summaries, the standard deviation will be presented to two decimal place greater than the original data, the mean and median will be presented to one decimal place greater than the original data and the minimum and maximum will be presented to the same number of decimal places as the original data.

For calculation of the proportion, one decimal place will be presented.

The rounding will be performed to the closest integer/first decimal using the common mid-point between the two consecutive values (e.g. 5.0 to 5.4 will be rounded to an integer of 5, and 5.5 to 5.9 will be rounded to an integer of 6)

## **Analysis Populations**

- The All subjects screened will include all subjects during screening evaluations.
- The Safety population will include all subjects who receive any amount of Alpha-1 MP.
- The PK population (GTI1401 only) will include all subjects who receive Alpha-1 MP dose and have sufficient samples to calculate the PK parameters.

### 5.6 Denominator

Unless otherwise mentioned, denominator of percentage in each table will be the number of population designated in each table.

# 6 Subject Disposition

| 6.1 Summary Table of Subject Disposition | | |
|---|---|---|
| Population | : | All subjects screened |
| Contents | : | The number of all subjects screened |
| | | • The number of all subjects dosed with Alpha-1 MP (Safety |
| | | population) |
| | | The number and percentage of all subjects in PK population |

| 6.2 Summary Table of Subjects Who Discontinue from the Study | | |
|---|---|---|
| Population | lation : Safety population | |
| Contents | : | • The number and percentage of subjects who complete the study |
| | | • The number and percentage of subjects who discontinue from the |
| | | study by reason for discontinuation |

Disposition status will be listed for all subjects. A listing will also be provided for screening failure subjects.

# 7 Protocol Deviations

| 7.1 Summary Table of Protocol Deviations | | |
|---|---|---|
| Population | : | Safety population |
| Contents | · | The number and percentage of deviations by type and severity will be summarized. Deviations from the protocol will be identified during the study and discussed in the data review meeting. Protocol deviation is defined in "GTI1401 and OLE Protocol Deviation Guidance_24Oct2016_Biling_Clean.pdf" Listing of all deviation. |

# 8 Demographics

| 8.1 Summary Table of Demographics | |
|---|---|
| Population | Safety population |
| Contents | For continuous variables, mean, standard deviation, median, and minimum/maximum will be provided. For categorical/qualitative data, frequency counts will be provided (For pregnancy status, the percentage of population is not included). Listing of following contests is provided separately. • Demographics (including alpha <sub>1</sub> - Antitrypsin Deficiency history) • Smoking history • Medical history |
| Analysis<br>variables | Contents, category and digit to be displayed are showed in the following table. |

| Contents | Category | Digits to be displayed |
|---|---|---|
| Sex | Male<br>Female | |
| Age [years] | | Integer |
| Race | Asian | |
| Weight [kg] | | 1 decimal place |
| Height [cm] | | 1 decimal place |
| Pregnancy status | NA (Males are included in this category) Negative Positive | |
| Smoking status | Never Former (>100 cigarettes or equivalent of tobacco in subject's lifetime) Current (not eligible for study) | |
| Total alpha <sub>1</sub> -PI serum level at time of diagnosis [mg/dL] | | 1 decimal place |
| Time since First Diagnosis of alpha <sub>1</sub> -Antitrypsin Deficiency [years] | | 1 decimal place |
| Best FEV <sub>1</sub> [L] at Baseline | | 2 decimal place |
| Best FVC [L] at Baseline | | 2 decimal place |
| FEV <sub>1</sub> Predicted [%] | 0=< < 30<br>30=< < 70<br>70=< <100 | |
| FEV <sub>1</sub> Predicted [%] | | 1 decimal place |

| Grifols Therapeutics Inc. | Statistical Analysis Plan |
|---------------------------|---------------------------|
| GTI1401/ GTI1401-OLE | 21MAR2017 |

| 15th Percentile of lung Density [g/L] | 1 decimal place |
|---------------------------------------|-----------------|
| Mean lung density [g/L] | 1 decimal place |

#### 9 Treatments and Medications

## 9.1 Prior and Concomitant Medications

Definition of prior medication and concomitant medication for GTI 1401 Prior medications are defined as any medication which ended before the first infusion of study drug of GTI 1401.

Concomitant medications are defined as any medication which is started on or after the first infusion of study drug of GTI 1401 or any medication taken prior to the first infusion of study drug of GTI 1401 and continued after the first infusion of study drug of GTI 1401.

### Definition concomitant medication for GTI 1401-OLE

Concomitant medications are defined as any medication which is started on or after the first infusion of study drug of GTI 1401-OLE or any medication taken prior to the first infusion of study drug of GTI 1401-OLE and continued after the first infusion of study drug of GTI 1401-OLE.

| 9.1.1 Summary Table of Prior and Concomitant Medication | | |
|---|---|---|
| Population | : | Safety population |
| Contents | •• | Summaries of all medications taken during the course of the study will be presented in tabular form and coded using ATC classification codes via the World Health Organization Drug classification Dictionary (WHO-DD). All medications will be summarized and sorted alphabetically by medication class (i.e., ATC level 2) and medication sub-class (i.e., ATC level 4). If the ATC level 4 term is missing, the ATC level 3 term will be used in the medication summary table and data listing. For the summary tables, if a subject has taken a concomitant medication more than once, the subject will be counted only once. |
| | | All medications will be listed by subject. New medications starting after the first infusion will be indicated if the medication start date relative to the first study drug infusion is greater than 0 in the subject data listing. |

## 9.2 Extent of Exposure

| 9.2.1 Summary Table of Drug Exposure | |
|--------------------------------------|----|
| Population : Safety populati | on |

| Contents | | Following contents regarding to exposure information are summarized. Digits to be displayed are showed in Table A Treatment duration [Week] Number of infusions received Total volume infused [mL] Volume infused per week [mL] Infusion duration [Minute] |
|---|---|---|
| | ŗ | Treatment duration in weeks is calculated as: |
| | | (The Last Dose Date – The First Dose Date + 7) / 7 |
| | , | Volume infused per week is calculated as: |
| | | the Total Volume Infused [mL] / the Treatment Duration [Week] |
| | ] | Infusion Duration is calculated as: |
| | | the Infusion Stop Time [HH:MM] —<br>the Infusion Start Time [HH:MM] + 1 |
| | | For Infusion Duration, the summary statistics will be calculated for mean duration of each week. |
| | | A list will be provided for Alpha-1 MP dose, volume prepared, and volume infused. |

# Table A:

| Contents | Digits to be displayed |
|------------------------------|------------------------|
| Treatment duration [week] | 1 decimal place |
| Number of infusions received | Integer |
| Total volume infused [mL] | 1 decimal place |
| Volume infused per week [mL] | 1 decimal place |
| Infusion duration [minute] | Integer |

| 9.2.2 Summary Table of Infusion Interruptions | | |
|---|---|---|
| Population | : | Safety population |
| Contents | : | The number and percentage of infusion with interruptions will be |
| | | summarized by analysis visit. |
| | | Reasons for interruptions will be displayed in the listings. |

## 9.3 Treatment Compliance

Treatment compliance will be calculated as:

$$\frac{\textit{Total Volume Infused}}{\textit{Total Volume Prepared}} \times 100\%$$

The total volume prepared is collected on the eCRF and is calculated based on the subject's weight at baseline.

The total volume prepared and dispensed by pharmacist is the intended dose volume a subject should be given based on the body weight.

Infusion compliance will be calculated as:

$$\frac{\textit{The Number of Actual Infusions}}{\textit{The Number of Infusions Expected}} \times 100\%$$

For subjects who drop out from the study early, the number of infusions expected will depend on the number of weeks the subjects are in the study.

| 9.3.1 Summa | ıry T | able of Treatment Compliance |
|---|---|---|
| Population | : | Safety population |
| Contents | • | <ul> <li>Following contents will be displayed.</li> <li>Summary of treatment compliance [%]</li> <li>The number of subjects with treatment compliance &gt;= 80%</li> <li>Summary of infusion compliance [%]</li> <li>A listing of treatment compliance will be provided.</li> </ul> |

### 10 Exploratory Analysis

## 10.1 PK Analysis (GTI1401 only)

Alpha<sub>1</sub>-Proteinase Inhibitor (alpha<sub>1</sub>-PI) concentrations in serum will be measured by validated content assay. The concentration data will be presented and summarized. Time points recorded on CRF will be used as analysis time points.

Time Table for Week 8 and Week 9

| | Actual elapsed | Nominal time point | |
|-------|----------------|--------------------|----------------------|
| Visit | time | (numeric version) | Scheduled time point |
| | (real-time) | (hours) | |

| Visit | Actual elapsed time (real-time) | Nominal time point (numeric version) (hours) | Scheduled time point |
|---|---|---|---|
| Week 8 | 0 | 0 | Immediately before the intravenous infusion |
| Week 8 | 0.30 | 0.25 | Immediately after the intravenous infusion (after flushing the infusion line with physiological saline) (at 0 hours) |
| Week 8 | 0.55 | 0.5 | 15 minutes after completion of the intravenous infusion |
| Week 8 | 2.35 | 2.25 | 2 hours after completion of the intravenous infusion |
| Week 8 | 4.67 | 4.25 | 4 hours after completion of the intravenous infusion |
| Week 8 | 8.67 | 8.25 | 8 hours after completion of the intravenous infusion |
| Week 8 | 26.02 | 24.25 | 24 ± 4 hours (1 day after completion of the intravenous infusion) |
| Week 8 | 49.17 | 48.25 | 48 ± 4 hours (2 days after completion of the intravenous infusion) |
| Week 8 | 120.58 | 120.25 | 120 hours ± 1 day (5 days after completion of the intravenous infusion) |
| Week 9 | 169.50 | 168.25 | 168 hours ± 1 day (7 days<br>after completion of the<br>intravenous infusion)<br>(Week 9) |

| 10.1.1 Sumn | nary [ | Table of Alpha <sub>1</sub> -PI Concentrations |
|---|---|---|
| Population | : | PK population |
| Contents | ÷ | Alpha <sub>1</sub> -PI concentrations will be summarized. The summaries will include n, mean (SD), coefficient of variation (%CV) (=SD/Arithmetic mean), median, minimum, maximum as well as geometric mean. |
| Digit | : | 2 decimal places will be displayed for summary table of alpha <sub>1</sub> -PI Concentrations. |
| Analysis | : | Immediately before the intravenous infusion |

| visit | <ul> <li>Immediately after infusion completion (after sodium chloride [NaCl] flush) (0 hour)</li> <li>15 minutes after infusion completion</li> <li>2 hours after infusion completion</li> <li>4 hours after infusion completion</li> <li>8 hours after infusion completion</li> <li>24±4 hours (1 day after infusion completion)</li> <li>48±4 hours (2 days after infusion completion)</li> <li>120 hours ± 1 day (5 days after infusion completion)</li> <li>168 hours ± 1 day (7 days after infusion completion) (Week 9 Visit)</li> <li>Serum concentrations of alpha<sub>1</sub>-PI determined by content assay will be presented in a listing by subject, study week, and scheduled or nominal time point.</li> </ul> |
|---|---|
| | This data listing will provide details of all planned plasma collection time points (scheduled and nominal times as specified in Section 12.1), actual collection date and clock times and elapsed times from the start of the study drug infusion, as well as alpha <sub>1</sub> -PI concentrations. Samples excluded from PK analysis will be flagged. |
| | The date/clock time for the start and completion of study drug infusion, the actual volume infused, and the actual dose infused (mg/kg) at Week 8 (PK assessment visit) will be presented in a separate listing. |

| 10.1.2 Sumn | nary ' | Table of Trough (pre-infusion) Levels (C <sub>min</sub> ) and mean C <sub>min</sub> |
|---|---|---|
| Population | : | PK population |
| Contents : | | <ul> <li>This table include following contents.</li> <li>Summary of trough (pre-infusion) levels (C<sub>min</sub>) and mean C<sub>min</sub> at steady state by week number (for C<sub>min</sub>).</li> <li>Mean C<sub>min</sub> calculated by the trough levels from weeks 7, 8, and 9 (exclude Week 1).</li> </ul> |
| | | • Number and Proportion with mean $C_{min}$ of alpha <sub>1</sub> -PI Concentration >= 50 mg/dL (=11.3 $\mu$ M nearly equal to 11 $\mu$ M which is defined in ATS/ERS statement in 2003). A conversion factor of 0.226 based on the protein only molecular weight of 44.3 KDa for alpha <sub>1</sub> -PI is used for converting mg/dL to $\mu$ M (i.e., 1 mg/dL alpha <sub>1</sub> -PI = 0.226 $\mu$ M). |
| | | No data imputations will be involved in the above concentration data listings, summaries, or figures. |
| | | Trough (pre-infusion) levels (C <sub>min</sub> ) and mean C <sub>min</sub> at steady state will |

| | | be listed |
|---|---|---|
| Digit | : | 2 decimal places will be displayed for summary table of C <sub>min</sub> . |
| Analysis | : | Week 1, Week 7, Week 8 and Week 9, |
| visit (only | | *mean $C_{min}$ = Average of $C_{min}$ of each patient measured at Week 7, |
| C <sub>min</sub> ) | | Week 8 and Week 9 (exclude Week 1) |

| 10.1.3 Figures of Concentration Versus Time Curves of Individual Subjects | | |
|---|---|---|
| Population | n : PK population | |
| Contents | : | For concentration data, serum alpha <sub>1</sub> -PI concentration versus time |
| | | curves following 8 weeks of treatments in individual subjects will be |
| | | presented in one figure with the actual elapsed time from the start of |
| | | the study drug infusion plotted on the x-axis. |

| 10.1.4 Figures of Concentration Versus Time Curves of All Subjects | | |
|---|---|---|
| Population | : | PK population |
| Contents | • | For all subjects combined, mean or median plasma alpha <sub>1</sub> -PI concentration versus time curves following 8 weeks of treatments will be presented in one figure with the nominal time plotted on the x-axis. |

All serum alpha<sub>1</sub>-PI concentration vs. time curves will be plotted on both linear and semilog scales.

A spaghetti plot (on the linear scale only) will be presented for all subjects following 8 weeks of treatment for concentration values vs nominal time.

#### Calculation of PK Parameters

The pharmacokinetic profiles of alpha<sub>1</sub>-PI following weekly administration of Alpha-1 MP will be characterized by pharmacokinetic parameters, including area under the curve (AUC) at steady state following 8 weeks of weekly infusions (AUC<sub>0-7days</sub>), maximum concentration ( $C_{max}$ ), time to first observed maximum concentration ( $t_{max}$ ), and half-life ( $t_{1/2}$ ), based on alpha<sub>1</sub>-PI concentrations in serum measured using content assay.

All PK parameters will be calculated using non-compartmental methods with WinNonlin software (Pharsight Corporation, Cary NC).

The pharmacokinetic parameters of interest are determined as follows:

| $AUC_{0-7days}$ | area und | er the | conce | ntration | vs. 1 | time o | curve a | at stea | dy state | over | the |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | _ | | | | | | |

weekly dosing interval (time 0 to 7 days), calculated by a combination of linear and logarithmic trapezoidal methods and expressed in the unit of concentration x time (mg·hr/dL). The linear trapezoidal method will be used for all incremental trapezoids arising from increasing concentrations and the logarithmic trapezoidal method will be used for those arising from

decreasing concentrations.

C<sub>max</sub> the first observed peak serum alpha<sub>1</sub>-PI concentration following drug infusion obtained directly from the experimental data without

interpolation, expressed in concentration units (mg/dL).

t<sub>max</sub> the observed time to reach peak serum alpha<sub>1</sub>-PI concentration obtained directly from the experimental data without interpolation,

expressed in time units (hour). If there are more than one maximum observed concentration, the  $t_{\text{max}}$  is the time to the first

observed peak concentration.

 $t_{1/2}$  the terminal half-life, calculated as  $(ln2)/K_{el}$ , expressed in time

units (hour). The apparent terminal first-order elimination rate constant, determined by linear regression analysis of the natural log-linear segment of the plasma concentration-time curve, expressed in time<sup>-1</sup> units (1/hour). At least 3 time points over 7 days following the treatment at week 8 will be included in the determination of K<sub>el</sub> (Points prior to Cmax or prior to the end of

infusion are not used).

C<sub>min</sub> the observed serum concentrations prior to the start of infusions obtained at Weeks 7, 8 and at 7 days (168 hours) post infusion at

Week 8, expressed in concentration units (mg/dL).

Mean C<sub>min</sub>

the average trough concentration at steady state, calculated as the mean value using the three  $C_{min}$  measurements obtained at Weeks 7, 8 and at 7 days (168 hours) post infusion at Week 9.

## Analysis of PK Parameters

For PK parameters descriptive statistics and geometric mean (except t<sub>max</sub>) will be calculated.

| 10.1.5 Summary of PK Parameters | | |
|---|---|---|
| Population | : | PK population |
| Contents | • | For following PK parameters, descriptive statistics including n, mean, standard deviation (SD), %CV, median, minimum, maximum and geometric mean (except t <sub>max</sub> ) will be calculated. The digits to be displayed and units will be described in Table B. Data listing for PK parameter will be provided. |

#### Table B

| Contents | Digits to be displayed |
|-----------------------------|------------------------|
| $AUC_{0-7days}$ [mg·hr/dL)] | 1 decimal place |
| $C_{max}[mg/dL]$ | 2 decimal place |
| t <sub>max</sub> [hours] | 2 decimal place |
| t <sub>1/2</sub> [hours] | 2 decimal place |

### 10.2 Lung density

Subjects will undergo CT scanning for diagnosis of clinically apparent pulmonary emphysema in GTI1401 study. This CT scan data will also serve as the baseline measurement of lung density for GTI1401-OLE study. Lung density collected by the CT scan data will be summarized in Demographics (parameter name=both).

In GTI1401-OLE study, the CT scan will be performed and summarized at Ext Week 52. The CT scan data will be accumulated for the future evaluation of lung density.

| 10.2.1 Summ | nary | Table of Lung Density |
|---|---|---|
| Population | : | Safety population |
| Contents | • | For following parameters and locations, descriptive statistics including n, mean, standard deviation (SD), %CV, median, minimum and maximum will be calculated. The digits to be displayed, units and all locaion will be described in Table: Lung Density Parameter and Table: Target Location. Data listing for Lung density parameters will be provided. |

Table: Lung Density Parameter

| Contents | Conversion formula for analysis value | Digits to be displayed |
|---|---|---|
| Hu value 15 percentile [g/L] | Original value [housfield unit] + 1000 | 1 decimal place |
| Mean [g/L] | Original value [housfield unit] + 1000 | 1 decimal place |
| Standard deviation [g/L] | Original value [housfield unit] + 1000 | 1 decimal place |
| Percent below -856 hu [%] | Original value | 1 decimal place |
| Percent below -910 hu [%] | Original value | 1 decimal place |
| Percent below -950 hu [%] | Original value | 1 decimal place |
| Total volume in cm3 [mL] | Original value | 1 decimal place |
| Air volume in cm3 [mL] | Original value | 1 decimal place |

Table: Target Location

| 1 401 | | Tuiget Docution |
|-------|---|---------------------------|
| 1 | : | Lung |
| 2 | : | Lung, Left |
| 3 | : | Lung, Left Lower Lobe |
| 4 | : | Lung, Left Upper Lobe |
| 5 | : | Lung, Right |
| 6 | : | Lung, Right Lower Lobe |
| 7 | : | Lung, Right Middle Lobe |
| 8 | : | Lung, Right Upper Lobe |
| 9 | : | Lung, Thirds Left Lower |
| 10 | : | Lung, Thirds Left Middle |
| 11 | : | Lung, Thirds Left Upper |
| 12 | : | Lung, Thirds Right Lower |
| 13 | : | Lung, Thirds Right Middle |
| 14 | : | Lung, Thirds Right Upper |

# 11 Safety Analysis

# 11.1 Adverse Events

# **Definition of Adverse Events**

| Adverse Event: | An AE is any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. |
|---|---|
| | An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the IMP. |
| | In this protocol, non-serious COPD exacerbation will not be considered as adverse events unless SAE. |
| TEAE for GTI 1401 | Treatment emergent adverse events (TEAE) for GTI 1401 will defined as any adverse event occurred after or on the first study drug infusion of GTI 1401 to the final visit of GTI 1401. |
| | For any subject, all AEs that occur at any time from the beginning of Alpha-1 MP administration until the final visit of the clinical trial will be considered as TEAE. |
| | All tables regarding to Adverse Events are restricted to TEAE. |
| TEAE for GTI1401-OLE | Treatment emergent adverse events (TEAE) for GTI 1401-OLE will defined as any adverse event occurred after or on the first study drug infusion of GTI 1401-OLE to the final visit of GTI 1401-OLE or adverse event which continue from GTI 1401 to GTI 1401-OLE. |
| | For any subject, all AEs that occur at any time from the beginning of Alpha-1 MP administration until the final visit of the clinical trial will be considered as TEAEs |
| | All tables regarding to Adverse Events are restricted to TEAE. |
| Adverse Drug Reaction (ADR): | The phrase "responses to a medicinal product" means that a causal relationship between a medicinal product or study treatment and an AE is at least a reasonable possibility, that is, the relationship cannot be ruled out. |

| | When an AE is classified, assessing causal relationship by the Investigator, as "definitive", "probable", "possible" or "doubtful/unlikely", the event will be defined as a suspected ADR. When the causal relationship is labeled "Unrelated", then it will be considered that the AE is not imputable to the study treatment and it is not a suspected ADR. |
|---|---|
| Serious Adverse Events (SAEs): | Any event reported on the AE CRF form with the serious field ticked "Yes". |
| | A SAE is any untoward medical occurrence that at any dose: |
| | Results in death |
| | Is life-threatening |
| | Note: The term "life-threatening" in this definition refers to an event in which the subject is at risk of death at the time of the event; it does not refer to an event that hypothetically might cause death if it were more severe. |
| | Requires inpatient hospitalization or prolongation of existing hospitalization |
| | Results in persistent or significant disability/incapacity |
| | Is a congenital anomaly/birth defect |
| Events of Special Interest: | Events of special interest include the following: All COPD exacerbations occurring during the study will be recorded. Each subject will be assessed for signs and symptoms of exacerbations at each study visit as specified in Appendix 1 and Appendix 2. Given that COPD exacerbations are part of the natural history of AATD, COPD exacerbations will not be reported as AEs unless a COPD exacerbation meets the criteria of a SAE. If an exacerbation meets criteria for a SAE, it will be reported as such, and the standard of care should be followed. Results from standard of care should be obtained and reported. |

Adverse events with incomplete start dates will be considered treatment emergent (TEAE) if:

• Day and Month are missing and the year is equal to or after the year of the first study drug dose date of each study (1401/1401-OLE);

- Day is missing, month is present and the month is equal or after the month of first dose of each study (1401/1401-OLE) and the year is equal or after the year of first dose date of each study (1401/1401-OLE);
- Day is missing and the year is equal to the year of the first infusion date of each study (1401/1401-OLE) and the month is equal to or after the month of the first infusion date of each study (1401/1401-OLE);
- Complete date is missing.

The AE tables will include the number and percentage of subjects by MedDRA primary System Organ Classes (SOC) - sorted by alphabetical order, MedDRA Preferred Terms (PT) - sorted by alphabetical order. A subject with more than one occurrence of the same adverse event in a particular system organ class/preferred term will be counted only once in the total of those experiencing adverse events in that particular system organ class/preferred term.

If a subject experiences the same adverse event at more than one severity, or with more than one relationship to study drug, the most severe rating or the stronger causal relationship to study drug will be given precedence. Any missing severity/relationship will be accounted as "worst case" as related in the tables.

All AE tables will be provided without separating AE occurred during treatment period with Follow-up period.

| 11.1.1 Overv | 11.1.1 Overview of AEs | |
|---|---|---|
| Population | : | Safety population |
| Contents | • | Overview AE table will be tabulated and will present number and percentages of subjects and number of events with following items. |
| | | <ul> <li>AEs</li> <li>ADRs</li> <li>AEs with fatal outcome</li> <li>SAEs</li> <li>AEs leading to premature discontinuation from the study</li> <li>Events of special interest</li> </ul> |

| 11.1.2 Summary Table of AEs ADRs | | |
|---|---|---|
| 11.1.3 Summ | 11.1.3 Summary Table of ADRs | |
| Population | : | Safety population |
| Contents | : | The number and percentage of incidences of AEs and ADRs in separate table by SOC and PT |

## 11.1.3 Summary Table of AEs by Causality

| Grifols Therapeutics Inc. | Statistical Analysis Plan |
|---------------------------|---------------------------|
| GTI1401/ GTI1401-OLE | 21MAR2017 |

| Population | : | Safety population |
|---|---|---|
| Contents | : | The number and percentage of incidences of AEs by causality based |
| | | on SOC and PT |

| 11.1.4 Summary Table of AEs by Severity | | |
|---|---|---|
| 11.1.5 Summary Table of ADRs by Severity | | |
| Population | : | Safety population |
| Contents | : | The number and percentage of incidences of AEs, and ADRs by |
| | | severity based on SOC and PT will be summarized. |

Following Listings regarding AEs will be provided.

- AEs
- SAEs
- Subjects with deaths
- AEs leading to premature discontinuation from the study AEs with Non-Serious COPD Exacerbation

# 11.2 Laboratory Tests

| 11.2.1 Summary Table of Laboratory Test | | |
|---|---|---|
| Population | : | Safety population |
| Contents | • | Summary statistics for original value and change from Baseline will be provided The analysis variables are defined in appendix for laboratory parameter. For Laboratory results, a data listing will be provided. |
| Analysis<br>Visit for<br>1401 | • | Baseline, Week 5, Week 9 |
| Analysis<br>Visit for<br>1401- OLE | : | Baseline, Ext Week 26, Ext Week 52 |

| 11.2.2 Summary Shift Table of Laboratory Test (Low, Normal and High) | | |
|---|---|---|
| 11.2.3 Summ | nary | Shift Table of Laboratory Test (Normal and Abnormal) |
| Population | Population : Safety population | |
| Contents | : | Shift tables for laboratory test with normal range will be provided. The analysis variables are defined in appendix for laboratory parameter |
| Analysis<br>Visit for | : | Baseline, Week 5, Week 9 |

| Grifols Therapeutics Inc. | Statistical Analysis Plan |
|---------------------------|---------------------------|
| GTI1401/ GTI1401-OLE | 21MAR2017 |

| 1401 | | |
|-----------|---|------------------------------------|
| Analysis | : | Baseline, Ext Week 26, Ext Week 52 |
| Visit for | | |
| 1401- OLE | | |

# 11.3 Vital Signs

| 11.3.1 Sumn | nary ' | Table of Vital Signs |
|---|---|---|
| Population | : | Safety population |
| Contents | · | Summary statistics for original value and change from Baseline will be provided. The analysis variables are displayed in Table C. For vital signs results, a data listing will be provided. |
| Analysis<br>Visit for<br>1401 | : | Week 1 prior to Infusion (Baseline) and Week 1 (After completion of infusion), Week 2 ~ Week 8 (Prior to infusion / After completion of infusion) |
| Analysis<br>Visit for<br>1401- OLE | : | Week 1 prior to Infusion (Baseline), Ext Week 1 ~ Ext Week 52 (Prior to infusion / After completion of infusion ) |

# Table C:

| Contents | Digits to be displayed |
|---------------------------------------|------------------------|
| Pulse rate [BEATS/MIN] | Integer |
| Systolic blood pressure [mmHg] | Integer |
| Diastolic blood pressure [mmHg] | |
| Body temperature [C] | 1 decimal place |
| Respiratory rate [breaths per minute] | Integer |

# 11.4 Electrocardiogram

| 11.4.1 Summary Table of Electrocardiogram | | |
|---|---|---|
| Population | : | Safety population |
| Contents | • | Shift tables for electrocardiogram will be provided. The analysis variables are displayed in Table D. For electrocardiogram results, a data listing will be provided. |
| Analysis<br>Visit for<br>1401 | • | Baseline, Week 9 |
| Analysis<br>Visit for<br>1401-OLE | : | Baseline, Ext Week 26, Ext Week 52 |

# Table D:

| Contents | Category |
|-------------------|----------|
| Electrocardiogram | Normal |
| | Abnormal |

# 11.5 Urine Cotinine Test

| 11.5.1 Summary Table of Urine Cotinine Tests | | |
|---|---|---|
| Population | : | Safety population |
| Contents | : | Shift table will be provided for Baseline value and the change from Baseline. The analysis variables are displayed in Table E. |
| Analysis<br>Visit for<br>1401 | : | Baseline, Week 5, Week 9 |
| Analysis<br>Visit for<br>1401-OLE | : | Baseline, Ext Week 26, Ext Week 52 |

# Table E:

| Contents | Category |
|-----------------------|----------|
| Urine cotinine result | Negative |
| | Positive |

# 11.6 Pulmonary Function Tests

| 11.6.1 Sumn | 11.6.1 Summary Table of Pulmonary Function Tests (FEV <sub>1</sub> and FVC) | |
|---|---|---|
| Population | : | Safety population |
| Contents | : | Summary statistics for original value and change from Baseline value will be provided for both "PRE-BRONCHODILATOR" and "POST-BRONCHODILATOR" separately. The analysis variables are displayed in Table F. |
| Analysis<br>Visit for<br>1401 | • | Screening, (Baseline), Week 5, Week 9 |
| Analysis<br>Visit for<br>1401-OLE | • | Screening (Baeline), Ext Week 26, Ext Week 52 |

| 11.6.2 Summary Table of Pulmonary Function Tests (FEV <sub>1</sub> % Predicted) | | |
|---|---|---|
| Population | : | Safety population |
| Contents | : | Frequency counts and summary statistics will be provided for both "PRE-BRONCHODILATOR" and "POST-BRONCHODILATOR" separately. The analysis variables are displayed in Table F. |
| Analysis<br>Visit for<br>1401 | ÷ | Screening, (Baseline), Week 5, Week 9 |
| Analysis<br>Visit for<br>1401-OLE | : | Screening (Baeline), Ext Week 26, Ext Week 52 |

# Table F:

| Contents | Digits to be displayed |
|-----------------------------------------|------------------------------------|
| Best FEV <sub>1</sub> [L] | 2 decimal place |
| Best FVC [L] | 2 decimal place |
| FEV <sub>1</sub> predicted [%] | Integer |
| FEV <sub>1</sub> predicted [%] category | 0=< < 30 |
| | 0=< < 30<br>30=< < 70<br>70=< <100 |
| | 70=<<100 |

For Pulmonary Function Tests, a data listing will be provided.

# 11.7 Pregnancy Tests

For pregnancy test, a data listing will be provided.

## 11.8 CT Scan

For CT Scan (densitometry), a data listing including lung density will be provided.

# 11.9 Physical Examination

For physical examination, a data listing will be provided.

# 12 Interim Analysis

No interim analysis is planned.

# 13 Changes in Planned Analysis

There are no changes in the planned analysis.

# **Appendix 1** Schedule of Study Procedures – GTI1401

| Trial period | Screening | Treatment <sup>a</sup> | | | | | | | | | | | Follow-up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit <sup>a</sup> | Day -21 to<br>the day<br>before<br>Week1 | Week 1<br>(baseline) | Week 2 | Week3 | Week 4 | Week 5 | Week 6 | Week 7 | Week 8 | PK1 | PK2 | PK5 | Week 9<br>(Study completion) <sup>b</sup> | Week 12<br>(Study<br>completion) <sup>c</sup> |
| Informed consent | X | | | | | | | | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | | | | | | | | |
| Assignment of subject number | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Age, sex | X | | | | | | | | | | | | | |
| CT Scan (densitometry) | $X^d$ | | | | | | | | | | | | | |
| Physical examination<br>(excluding breast and urogenital examination) | X | | | | | | | | | | | | X | X |
| Body height | X | | | | | | | | | | | | | |
| Body weight | X | Xe | | | | Xe | | | | | | | | |
| Blood sampling for viral safety assessment <sup>f</sup> | | X | | | | | | | | | | | | |
| Urine pregnancy test<br>(Only in women of childbearing potential) | X | | | | | X | | | | | | | X | X |
| Urinary cotinine level | X | | | | | X | | | | | | | X | X |
| Blood and urine sampling for laboratory tests<br>(Hematology, blood chemistry, urinalysis) | X | X <sup>g</sup> | | | | X <sup>g</sup> | | | | | | | X | X |
| Vital signs (Pulse rate, blood pressure, respiratory rate, body temperature) <sup>h</sup> | | X | X | X | X | X | X | X | X | | | | Х | X |
| 12-lead ECG | X | X | | | | | | | | | | | (X) | |
| Pulmonary function tests before and after administration of a bronchodilator (FEV $_{\rm l}$ and FVC) $^{\rm i}$ | X i | | | | | X i | | | | | | | X i | X i |
| Blood sampling for alpha <sub>1</sub> -PI concentration measurement | X <sup>j</sup> | X <sup>g</sup> | | | | | | X g | X k | X k | X k | X k | X k | |
| Intravenous infusion of Alpha-1 MP <sup>1</sup> | | X | X | X | X | X | X | X | X | | | | | |
| Observation of subjects after infusion of Alpha-1 MP <sup>m</sup> | | X | X | X | X | X | X | X | X | | | | | |
| Evaluation of COPD exacerbations | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Evaluation of adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Evaluation of concomitant medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
- a: The date of individual visits will be determined in relation to the date of the Week 1 (baseline) visit. The date of all visits after the screening visit and the Week 1 (baseline) visit will be arranged within a time window of ± 1 day. The PK evaluation period will start at the Week 8 visit and end at the Week 9 visit.
- b: At the Week 9 visit, subjects will be asked whether or not they would like to enter the extension trial (GTI1401-OLE). For subjects eligible for participation in the extension trial, the Week 9 visit will be the study completion visit for this clinical trial (GTI1401).
- c: Subjects not entering the extension trial (GTI1401-OLE) and subjects who receive Alpha-1 MP at any dose and discontinue this clinical trial early will be asked to return to the study center for the follow-up/study completion procedures and evaluations scheduled at the Week 12 visit. This visit should be made at the timing as close as possible to 4 weeks (i.e., 30 days) after the last dose of the investigational drug in the subject.
- d: CT densitometry scan should be performed anytime from the Screening Visit to the Week 1 (Baseline) Visit; if the CT densitometry scan is performed at the Week 1 (Baseline) Visit, then it must be performed prior to the first Alpha-1 MP infusion. This CT scan will measure lung density.
- e: Body weight will be used to calculate the Alpha-1 MP dose, and this recorded body weight will be used for dose calculation until the next scheduled body weight measurement.
- f: Blood samples for viral safety assessment (viral NAT and viral serologic test) will be collected before the intravenous infusions of Alpha-1 MP at the Week 1 (baseline) visit. However, the collected samples will be tested only if the subject shows clinical signs or symptoms suggestive of viral infection during the trial period. Only in this case will additional blood samples for viral NAT and viral serologic test be collected. All these collected blood samples will be stored until completion of all the tests in this clinical trial (GTI1401) and the extension trial (GTI1401-OLE).
- g: Sampling will be performed before each intravenous infusion of Alpha-1 MP.
- h: Vital signs will be checked immediately before and after each intravenous infusion of Alpha-1 MP.
- i: Pulmonary function tests after administration of a bronchodilator will be performed 15 to 30 minutes after administration of a bronchodilator. For a short-acting bronchodilator, subjects will receive 4 puffs of salbutamol given by an MDI and spacer in each pulmonary function testing. The same bronchodilator as that used at the start of the trial should be used throughout the trial period.
- j: Sampling will be performed in subjects with no previously documented alpha1-PI levels as measured by nephelometry (if it is unknown whether the subject's alpha1-PI level is <50 mg/dL or not).

Grifols Therapeutics Inc.

GTI1401/GTI1401-OLE

Statistical Analysis Plan
21MAR2017

k: Sampling time points of PK samples: 1) Immediately before the intravenous infusion; 2) Immediately after the intravenous infusion (after flushing the infusion line with physiological saline) (at 0 hours); 3) At 15 minutes after completion of the intravenous infusion; 4) At 2 hours after completion of the intravenous infusion; 5) At 4 hours after completion of the intravenous infusion; 7) At 24 ± 4 hours (1 day after completion of the intravenous infusion); 8) At 48 ± 4 hours (2 days after completion of the intravenous infusion); 9) At 120 hours ± 1 day (5 days after completion of the intravenous infusion); and 10) At 168 hours ± 1 day (7 days after completion of the intravenous infusion) (Week 9).

1: Weekly intravenous infusions of 60 mg/kg of Alpha-1 MP will be given under the supervision of the investigator or a designated person at each study center.

# **Appendix 2** Schedule of Study Procedures – GTI1401-OLE

| | Screening/Ex | t Week 1 Visit | Weekly | | Bi-Annu | ıal Visits | End of Study<br>Follow-Up |
|---|---|---|---|---|---|---|---|
| Visits Procedures/Assessments | Screening <sup>a</sup> | Initiation of<br>Infusion | On-Site Infusion Visits (Ext Weeks 2 to 52) | Quarterly Visits<br>(Ext Weeks 12, 24, 36,<br>48) | Ext Week 26 | Ext Week 52 | Assessment <sup>b</sup> (via phone call) (Ext Week 53) |
| Informed consent | X | | | | | X | |
| Inclusion/exclusion criteria | X | | | | | | |
| Subject number confirmed | X | | | | | | |
| Weight | | | | X | | | |
| Collection of virus safety retain samples | | | | | | X | |
| Physical exam (excludes breast and genitourinary) | | | | | X | X | |
| Urine pregnancy test (potential child-bearing females only) | | | | | X | X | |
| Urine cotinine | | | | | X | X | |
| Blood for hematology and chemistry laboratory assessments | | | | | X | X | |
| Blood for retains for possible future testing | | | | | X | X | |
| Urinalysis | | | | | X | X | |
| Vital signs (heart rate, blood pressure, respiratory rate, and temperature) | | X | X | X | X | X | |
| Pre- and post-bronchodilator PFTs (FEV <sub>1</sub> and FVC) | | | | | X | X | |
| Blood for Alpha <sub>1</sub> -PI level | | | | X | | | |
| Alpha-1 MP IV infusion | | X | X | X | X | X | |
| COPD exacerbation assessment | | | | | X | X | X |
| Adverse event assessment | | | X | X | X | X | X |
| Concomitant medications assessment | | | X | X | X | X | X |

# Appendix for Laboratory Parameter:

| Display<br>order | Category for Lab<br>Test | LB parameter code | LB parameters (SI unit) | Digit to be displayed |
|---|---|---|---|---|
| 1 | HEMATOLOG<br>Y | HGB | Hemoglobin [g/L] | Integer |
| 2 | HEMATOLOG<br>Y | НСТ | Hematocrit [%] | 1 decimal place |
| 3 | HEMATOLOG<br>Y | PLAT | Platelets [10^9/L] | Integer |
| 4 | HEMATOLOG<br>Y | RBCH | Erythrocytes [10^12/L] | 2 decimal place |
| 5 | HEMATOLOG<br>Y | WBCH | Leukocytes [10^9/L] | 1 decimal place |
| 6 | HEMATOLOG<br>Y | NEUT | Neutrophils [%] | Integer |
| 7 | HEMATOLOG<br>Y | LYM | Lymphocytes [%] | 1 decimal place |
| 8 | HEMATOLOG<br>Y | MONO | Monocytes [%] | 1 decimal place |
| 9 | HEMATOLOG<br>Y | EOS | Eosinophils [%] | 1 decimal place |
| 10 | HEMATOLOG<br>Y | BASO | Basophils [%] | 1 decimal place |
| 11 | CHEMISTRY | SODIUM | Sodium [mmol/L] | Integer |
| 12 | CHEMISTRY | K | Potassium [mmol/L] | 1 decimal place |
| 13 | CHEMISTRY | CREAT | Creatinine [mg/dL] | 2 decimal place |
| 14 | CHEMISTRY | CA | Calcium [mg/dL] | 1 decimal place |
| 15 | CHEMISTRY | UREAN | Urea Nitrogen [mg/dL] | Integer |
| 16 | CHEMISTRY | BICARB | Bicarbonate [mmol/L] | 1 decimal place |
| 17 | CHEMISTRY | ALB | Albumin [g/L] | Integer |
| 18 | CHEMISTRY | AST | Aspartate Aminotransferase [IU/L] | Integer |
| 19 | CHEMISTRY | ALT | Alanine Aminotransferase [IU/L] | Integer |
| 20 | CHEMISTRY | ALP | Alkaline Phosphatase [IU/L] | Integer |
| 21 | CHEMISTRY | GLUCC | Glucose [mg/dL] | Integer |
| 22 | CHEMISTRY | PROTC | Protein [g/L] | Integer |
| 23 | CHEMISTRY | BILI | Bilirubin [mg/dL] | 1 decimal place |
| 24 | URINALYSIS | PH | рН | |
| 25 | URINALYSIS | PROT | Protein | |
| 26 | URINALYSIS | GLUC | Glucose | |
| 27 | URINALYSIS | OCCBLD | Occult Blood | |
| 28 | URINALYSIS | MUCTH<br>R | Mucous Threads | |

# Layout Plan

## GT11401

Protocol title: A Multi-Center, Open-Label Study to Evaluate the Safety and Pharmacokinetics of

Weekly Intravenous Infusions of Alphal-Proteinase Inhibitor (Human) in Japanese Subjects with

GTI1401-OLE

Protocol title:

A Multi-Center, Open-Label Study to Evaluate the Long-term Safety of Weekly Intravenous Infusions of Alphal-Proteinase Inhibitor (Human) in Japanese Subjects with Alphal Antitrypsin Deficiency

Study code:

Alpha-1 MP

Sponsor:

Grifols Therapeutics Inc.

79 TW Alexander Drive Research Triangle Park, NC 27709

LP status:

0.1V

Date:

21MAR2017

Approval:

Har 23,2017



Date

# Change Record

| Version No. | Date | Author | Description of changes (revisions and reasons) |
|---|---|---|---|
| V0.1 | 2016/5/25 | | Created 1st draft |
| V0.2 | 2016/12/2 | | Incorporated client's review of 1st draft |
| V0.3 | 2016/3/1 | | Incorporated client's review of 2nd draft and MW input |
| V1.0 | 2016/3/21 | | Removed review comment |

| No ID of TFL | Tittle of TFLs | Statistic | al Analysis Plan | Number of Table | GTI1401 | GTI1401-OLE | Remarks |
|---|---|---|---|---|---|---|---|
| | | | ii Aliaiysis i iali | Number of Table | | | Remains |
| 1 Disp-1<br>2 Disp-2 | 6.1 Summary Table of Analysis Population 6.2 Summary Table of Subjects Who Discontinue From the Study | 6 Subject Disposition | | | 0 | 0 | |
| | 6.3 Listing of Subject Disposition | | | | | 0 | "6.4 Listing of Screening Failures" will be based on this table layout. |
| 4 Devi-1 | 7.1 Summary Table of Protocol Deviations | 7 Protocol Deviations | | | ŏ | <del>0</del> | 0.4 Eisting of Screening Failures will be based on this table layout. |
| | 7.2 Listing of Protocol Deviation | / Frotocol Deviations | | | ŏ | ŏ | |
| | | 8 Demographics | | | Ō | Ō | |
| | 8.2 Listing of Demographic Characteristics | | | | | 0 | |
| | 8.3 Listing of Smoking History | | | | 0 | 0 | |
| | 8.4 Listing of Medical History | | | | | 0 | WALL OF THE CO. T. L. |
| | • | 9 Treatments and Medications | 9.1 Prior and Concomitant Medication | | 0 | _ | "9.1.2 Summary Table of Concomitant Medication" will be based on this table layout |
| | 9.1.3 Listing of Medications | | 0.00 | | 0 | 0 | |
| 10 Exp-1 | 9.2.1 Summary Table of Drug Exposure 9.2.2 Summary Table of Infusion Interruptions | | 9.2 Extent of Exposure | | | 0 | |
| 11 Exp-2 | | | | | 0 | 0 | |
| 12 Exp-L1<br>13 Comp-1 | 9.2.3 Listing of Exposure Information 9.3.1 Summary Table of Treatment Compliance | | 0.27 | | 0 | 0 | |
| | 9.3.2 Listing of Treatment Compliance | | 9.3 Treatment Compliance | | 0 | 0 | |
| 15 Pk-1 | 10.1.1 Summary Table of Alpha1-PI Concentrations | 10 Exploratory Analysis | 10.1 PK Analysis (GTI1401 only) | | 0 | 0 | |
| 16 Pk-2 | 10.1.2 Summary Table of Trough (pre-infusion) Levels (Cmin) and mean Cmi | | 10.1 PK Analysis (G111401 only) | | 0 | | |
| 17 Pk-3 | 10.1.3 Figures of Concentration Versus Time Curves of Individual Subjects | | | | 0 | | |
| 18 Pk-4 | 10.1.4 Figures of Concentration Versus Time Curves of All Subjects | | | | 0 | | |
| 19 Pk-5 | 10.1.5 Summary of PK Parameters | | | | 0 | | |
| 20 Pk-L1 | 10.1.6 Listing of Alpha1-PI Concentrations (Week 8 and 9) | | | | 0 | | |
| 20 Pk-L1<br>21 Pk-L2 | 10.1.6 Listing of Alpha1-PI Concentrations (week 8 and 9) | | | | 0 | | |
| | č . | | | | 0 | | |
| 22 Pk-L3 | 10.1.8 Listing of Trough (pre-infusion) levels (Cmin) and mean Cmin | | | | | | |
| 23 Pk-L4 | 10.1.9 Listing of PK Parameters | | | | 0 | | |
| 24 Mo-1 | 10.2.1 Summary Table of Lung Density | | | | | | |
| 25 Mo-L1<br>26 AE-1 | 10.2.2 Listing of Lung Density<br>11.1.1 Overview of AEs | 1100. | 11.1 Adverse Events | | 0 | 0 | |
| 26 AE-1<br>27 AE-2 | 11.1.1 Overview of AEs 11.1.2 Summary Table of AEs | 11 Safety Analysis | 11.1 Adverse Events | | | | "11.1.3 Summary Table of ADRs" will be based on this table layout. |
| 28 AE-3 | 11.1.4 Summary Table of AEs 11.1.4 Summary Table of AEs by Causality | | | | | 0 | 11.1.5 Summary Table of ADRS will be based on this table layout. |
| | | | | | | - | HILLO THE CAPPEL OF THE THEFT OF THE THEFT |
| 29 AE-4 | 11.1.5 Summary Table of AEs by Severity | | | | | | "11.1.6 Summary Table of ADRs by Severity" will be based on this table layout. "11.1.10 Listing of AEs leading to Premature Discontinuation from the Study" will be based on this table |
| 30 AE-L1 | 11.1.7 Listing of AEs | | | | 0 | 0 | "11.1.10 Listing of ALs leading to Premature Discontinuation from the Study" will be based on this table layout. |
| 31 AE-L2 | 11.1.8 Listing of Death | | | | 0 | 0 | iayout. |
| 31 AE-L2<br>32 AE-L3 | 11.1.8 Listing of Death 11.1.9 Listing of SAE | | | | 0 | 0 | |
| 32 AE-L3<br>33 AE-L4 | 11.1.19 Listing of SAE 11.1.11 Listing of Non-Serious COPD Exacerbation | | | | 0 | 0 | |
| 34 Lb-1 | 11.2.1 Summary Table of Laboratory Test | | 11.2 Laboratory Tests | | | | Tables for all the laboratory examination item described on SAP will be based on this table layout |
| 35 Lb-2 | 11.2.2 Summary Fable of Laboratory Test (Low, Normal and High) | | 11.2 Laudiatory rests | | 0 | | Chemistry and hematology laboratory parameter described on SAP will be based on this table layout. |
| 36 Lb-3 | 11.2.2 Summary Shift Table of Laboratory Test (Low, Normal and High) 11.2.3 Summary Shift Table of Laboratory Test (Normal and Abnormal | | | | | | Urine laboratory parameter described on SAP will be based on this table layout. |
| 37 Lb-L1 | 11.2.3 Summary Sinit Table of Laboratory Test (Normal and Abnormal | | | | 0 | Ö | orme mooratory parameter described on order with oc based on this table layout. |
| 38 Vs-1 | 11.3.1 Summary Table of Vital Signs | | 11.3 Vital Signs | | | 0 | |
| 39 Vs-L1 | 11.3.2 Listing of Vital Signs | | 11.5 - Indi Digita | | 0 | Ö | |
| 40 Ecg-1 | 11.4.1 Summary Table of Electrocardiogram | | 11.4 Electrocardiogram | | ŏ | ŏ | |
| 41 Ecg-L1 | 11.4.2 Listing of Electrocardiogram | | ĕ | | Ō | Ō | |
| 42 Ur-1 | 11.5.1 Summary Table of Urine Cotinine Test | | 11.5 Urine Cotinine Test | | | ŏ | |
| 43 Ur-L1 | 11.5.2 Listing of Urine Cotinine Test | | | | | 0 | |
| 44 Pul-1 | 11.6.1 Summary Table of Pulmonary Function Tests (FEV1 and FVC) | | 11.6 Pulmonary Function Tests | | 0 | 0 | |
| 45 Pul-2 | 11.6.2 Summary Table of Pulmonary Function Tests (FEV1 % Predicted) | | - | | | 0 | |
| 46 Pul-L1 | 11.6.3 Listing of Pulmonary Function Tests | | | | 0 | O | |
| 47 Pr-L1 | 11.7 Listing for Pregnancy Tests | | 11.7 Pregnancy Test | | | 0 | |
| 48 CT-L1 | 11.8 Listing for CT Scan | | 11.8 CT Scan | | 0 | 0 | |
| 49 PE-L1 | 11.9 Listing for Physical Examination | | 11.9 Physical Examination | | 0 | 0 | |

# General Setting

| documents should allow printing in A4 without changing the page setup of the ents. scape orientation is preferred, portrait is allowed. ttom, left, and right: 2.54 cm (1 in) New Roman 9pt or larger for all tables, when space is an issue (i.e. in terms of the page setup), the following ns can be used (in the following order shown below): ing, abbreviation; |
|---|
| ents. scape orientation is preferred, portrait is allowed. ttom, left, and right: 2.54 cm (1 in) New Roman 9pt or larger for all tables, when space is an issue (i.e. in terms of the page setup), the following ns can be used (in the following order shown below): |
| ents. scape orientation is preferred, portrait is allowed. ttom, left, and right: 2.54 cm (1 in) New Roman 9pt or larger for all tables, when space is an issue (i.e. in terms of the page setup), the following ns can be used (in the following order shown below): |
| ttom, left, and right: 2.54 cm (1 in) New Roman 9pt or larger for all tables, when space is an issue (i.e. in terms of the page setup), the following ns can be used (in the following order shown below): |
| New Roman 9pt or larger for all tables, when space is an issue (i.e. in terms of the page setup), the following ns can be used (in the following order shown below): |
| tables, when space is an issue (i.e. in terms of the page setup), the following ns can be used (in the following order shown below): |
| ns can be used (in the following order shown below): |
| ables across pages; istings into sections. |
| oles, when there is no subject to be counted, '0' will be displayed. |
| case of percentage or summary statistics can not be calculated (e.g. Denominator there is no denominator), '-' will be displayed. If no subject to be counted and ninator >0 then display "0" instead of "0 (0.0)". |
| tput should be left aligned on the page. |
| and footnotes should be left aligned. |
| n headers and column contents for text variables should be left justified, while headers and column content for numeric variables should be centered. Senation of statistics, counts and percentages should be centered. |
| riables displayed as numerical output (including dates and concatenation of cs), and which have the same data format on all rows, the data should be aligned |
| decimal point and be centered within the column. |
| ( |

# General Setting for Title and Footnote

| Title1 | GTI 1401 | | | | | | Page 1 of x |
|---|---|---|---|---|---|---|---|
| Title2 | <x of="" section="" title=""></x> | | | | | | |
| Title3 | <pre><x of="" pre="" sect<="" sub="" title="" x=""></x></pre> | ion or title of table | e, listing and figure> | | | | |
| Title4 | <pre><x of="" pre="" table,<="" title="" x=""></x></pre> | listing and figure | > | | | | |
| Title5 | <target populaton=""></target> | | | | | | |
| | column1 | column2 | column3 | column4 | column5 | column6 | column7 |
| T 1 | . 11 6 | | | | | | |
| Footnote1 | table footnotes (if ne | | In this Layout Plan, | only the table for | otnotes will be | nresented | 1 |
| <br>E44 | table footnotes (if ne | | in each sheet. | omy the table for | othotes will be | presented | |
| Footnote n | table footnotes (if ne | | > For GTI1401-OLE, | title 1 will he cha | anged to "GTI1 | 4∩1-∩LF" | |
| Footnote n+1 | table footnotes (if ne | | , 101 G111 <del>1</del> 01-011, | THE I WILL BE CHE | inged to OIII. | | |
| Footnote n+2 | table footnotes (if ne | cessary) | | | | | - |

GTI 1401 6 Subject Disposition 6.1 Summary Table of Analysis Population

# All subjects screened

| Population | n (%) |
|-----------------------|---------|
| All subjects screened | XX |
| Safety population | XX |
| PK population | xx(xxx) |

<sup>\*</sup> Denominator of tabulation is the number of Safety Population

GTI 1401 6 Subject Disposition 6.2 Summary Table of Subjects Who Discontinue From the Study

| | N=88 |
|----------------------------------------------|-----------|
| Reason of Study Discontinuation | n (%) |
| Subjects who complete the study | xx (xx x) |
| Subjects who discontinue from the study | xx (xx x) |
| Adverse Event | xx (xx x) |
| Withdrawal By Subject (Does not Include AEs) | xx (xx x) |
| •••• | xx (xx x) |

<sup>\*</sup> Denominator of tabulation is the number of Safety Population

GTI 1401 6 Subject Disposition 6.3 Listing of Subject Disposition

# All subjects screened

| | | Date of | | | | |
|---|---|---|---|---|---|---|
| | | Screening /Date | | | | |
| | Safety/ | of Last Visit | Complete | Reason for Early | Reason for Exclusion of | Safety Reason for Exclusion of PK |
| Subject Number | PK Population | on (Study Day) | Study | Discontinuation | Population | Population |
| XXX | Y/N | yyyy-mm-dd / | N | | | |
| | | yyyy-mm-dd | | OTHER: xxx | | XXX |
| XXX | Y/Y | yyyy-mm-dd / | Y | | | |
| | | yyyy-mm-dd | | | | |
| XXX | | | | | | |

>Listing for "Screening Failures" will be also provided in same format. >Row 6 Column 3 will be changed to "Screening Failures".

>Sort order; Subject Number

>Date of last date for who completes study is date of completion of disposition event. Date of last date for who discontinues is date of discontinuation of disposition event.

GTI 1401 7 Protocol Deviations 7.1 Summary Table of Protocol Deviations

# Safety Population

| | | _ | _ | N | 1=88 | |
|---|---|---|---|---|---|---|
| | | | Critical | Major | Minor | Total |
| | | Reason of Protocol Deviation | n (%) | n (%) | n (%) | n (%) |
| Protocol deviation | No | | xx (xx.x) | xx (xx x) | xx (xx.x) | xx (xx x) |
| | Yes | | xx (xx.x) | xx (xx x) | xx (xx.x) | xx (xx x) |
| | | Entry Criteria | xx (xx.x) | xx (xx x) | xx (xx.x) | xx (xx x) |
| | | Investigational Product<br>Visit Schedule Criteria<br>Informed Consent | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx x)<br>xx (xx x)<br>xx (xx x) | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) | xx (xx x)<br>xx (xx x)<br>xx (xx x) |
| | | Conc. Medications | xx(xx.x)<br>xx(xx.x) | xx(xxx) | xx(xx.x) | xx(xxx) |
| | | Study Procedures | xx(xx.x) | xx (xx x) | xx (xx.x) | xx (xx x) |
| | | Laboratory / PK | xx (xx.x) | xx (xx x) | xx (xx.x) | xx (xx x) |
| | | Laboratory | xx(xx.x) | xx(xxx) | xx(xx.x) | xx(xxx) |

<sup>\*</sup> Denominator of tabulation is the number of Safety Population

>Only criteria which contain at least one subject will be displayed.

GTI 1401 7 Protocol Deviations 7.2 Listing of Protocol Deviation

# Safety Population

| | Subject | Category of Protocol | | |
|---|---|---|---|---|
| Site Name | Number | Deviation* | Severity | Details of Protocol Deviation |
| xxxxxxxxxx | XX | 1 | MAJOR | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XX | 2 | MINOR | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | XX | 1 | MAJOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxxxxxx | XX | 3 | MAJOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | XX | 1 | MAJOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxxxxxx | XX | 2 | MAJOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | XX | 4 | MAJOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | XX | 5 | MAJOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxxxxxx | XX | 5 | MAJOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | XX | 6 | MAJOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | xx | 7 | MINOR | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

<sup>\* 1.</sup> Entry Criteria 2. Investigational Product 3. Visit Schedule Criteria 4. Informed Consent 5. Conc. Medications 6. Study Procedures 7. Laboratory / PK 8. Laboratory

>Sort order;

Site, Subject Number, Category of Protocol Deviation

# 8 Demographics 8.1 Summary Table of Demographics

| | N=xx |
|-----------------------------------------|-------------|
| | n (%) |
| Sex | |
| Male | xx(xxx) |
| Female | xx (xx x) |
| Age [years] | |
| N | XX |
| Mean(S.D.) | xx x (xx.x) |
| Median | XX X |
| Min , Max | XX,XX |
| Race | |
| Asian | XX |
| Weight [kg] | |
| N | XX |
| Mean(S.D.) | xx x (xx.x) |
| Median | XX X |
| Min , Max | XX , XX |
| Height [cm] | |
| N | XX |
| Mean(S.D.) | xx x (xx.x) |
| Median | |
| Min , Max | XX , XX |
| Pregnancy status | |
| NA(Males are included in this category) | XX |
| Negative | XX |
| Positive | XX |

# 8 Demographics 8.1 Summary Table of Demographics

| | N=xx |
|---|---|
| | n (%) |
| Smoking status | XX |
| Never | XX |
| Former | XX |
| Current | |
| Total Alpha-1 serum level at time of diagnosis [mg/dL] | |
| N | XX |
| Mean(S.D.) | xx x (xx.x) |
| Median | XX X |
| Min, Max | XX , XX |
| Time since first diagnosis of Alpha-1 antitrypsin deficiency [years] *1 | |
| N | XX |
| Mean(S.D.) | xx x (xx.x) |
| Median | XX X |
| Min, Max | XX , XX |
| Best FEV1 [L] at Baseline for "PRE-BRONCHODILATOR" | xx |
| N | xx x (xx.x) |
| Mean(S.D.) | XX X |
| Median | XX,XX |
| Min , Max | |
| Best FVC [L] at Baseline for "PRE-BRONCHODILATOR" | xx |
| N | xx x (xx.x) |
| Mean(S.D.) | XX X |
| Median | XX,XX |
| Min, Max | |
| FEV1 predicted [%] for "PRE-BRONCHODILATOR" | xx |
| 0=<<30 | XX |
| 30=< < 70 | XX |
| 70=<<100 | |

# 8 Demographics 8.1 Summary Table of Demographics

| | N=xx |
|-----------------------------------------------------|-------------|
| | n (%) |
| Best FEV1 [L] at Baseline for "POST-BRONCHODILATOR" | xx |
| N | xx x (xx.x) |
| Mean(S.D.) | XX X |
| Median | XX , XX |
| Min , Max | , |
| Best FVC [L] at Baseline for "POST-BRONCHODILATOR" | xx |
| N | xx x (xx.x) |
| Mean(S.D.) | XX X |
| Median | XX,XX |
| Min , Max | |
| FEV1 predicted [%] for "POST-BRONCHODILATOR" | xx |
| 0=< < 30 | XX |
| 30=< < 70 | XX |
| 70=<<100 | |
| 15th Percentile of lung density [g/L] | |
| N | XX |
| Mean(S.D.) | xx x (xx.x) |
| Median | XX X |
| Min, Max | XX , XX |
| Mean lung density [g/L] | |
| N | XX |
| Mean(S.D.) | xx x (xx.x) |
| Median | XX X |
| Min, Max | XX,XX |

<sup>\*1</sup> Informed Consent Date - First Date of Diagnosis of Alpha-1 Antitrypsin Deficiency + 1 / 365

\* Denominator of tabulation is the number of Safety Population

GTI 1401 8 Demographics 8.2 Listing of Demographic Characteristics

Safety population

| | | | | | Total Alpha-1 | | | Emphysema | FEV1 [L] / Best FVC [L] at | FEV1 [L] / Best FVC [L] at |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | Serum Level | | | Diagnosed | Baseline for | Baseline for |
| | Sex/ | Weight | | | at Time of | | Date of Total | by CT Scan / | "PRE- | "POST- |
| Subject | Age/ | [kg]/ | Fertility Status/Birth | Smoking | Diagnosis | Date of First | Alpha-1 PI | Date of CT | BRONCHOD | BRONCHOD |
| Number | Race | Height [cm] | Control | Status | [mg/dL] | Diagnosis | Serum Level | scan | ILATOR" | ILATOR" |
| xx | xx /<br>xx / | xx /<br>xx | CHILDBEARING POTENTIAL /DOUBLE BARRIER METHODS | | xx | yyyy-mm-dd | yyyy-mm-dd | Y /<br>yyyy-mm-dd | | xx / xx |
| xx | Asian<br>xx /<br>xx /<br>xx | xx/<br>xx | SURGICALLY<br>STERILE | yyyy-mm-dd<br>NEVER | xx | yyyy-mm-dd | yyyy-mm-dd | N | | xx / xx |

>Sort order; Subject Number

8 Demographics

8.3 Listing of Smoking History

# Safety population

| Subject Number | Smoking History | Previous Smoking Type | Date of Last Smoking |
|---|---|---|---|
| XXXX | NEVER | | |
| | | CIGARS / | |
| xxxx | FORMER | PIPES | yyyy-mm-dd |
| | | CIGARS / | |
| XXXX | FORMER | CIGARETTES (xx x) | |

>Sort order; Subject Number

8 Demographics

8.4 Listing of Medical History

Safety population

# MedDRA System Organ

| Subject Number | Onset Date | Resolved Date | Class | Preferred Term | Verbatim Term |
|---|---|---|---|---|---|
| XXXX | yyyy-mm-dd | yyyy-mm-dd | XXXXXXXXX | уууууууу | ZZZZZZZZZ |
| | yyyy-mm-dd | ONGOING | XXXXXXXXX | уууууууу | ZZZZZZZZZ |
| XXXX | yyyy-mm-dd | yyyy-mm-dd | XXXXXXXXX | уууууууу | ZZZZZZZZZ |

>Sort order;

Subject Number, Onset Date, MedDRA System Organ Class, Preferred Term (Both alphabetical order)

- 9 Treatments and Medications
- 9.1 Prior and Concomitant Medications
- 9.1.1 Summary Table of Prior Medication

| | N=88 |
|---------------------------------------------|-----------|
| Who Drug ATC Term | n (%) |
| Subjects with at least one prior medication | xx (xx.x) |
| ATC2 | xx (xx.x) |
| ATC4 | xx (xx.x) |
| •••• | xx (xx.x) |
| ATC2 | xx (xx.x) |
| ATC4 | xx (xx.x) |
| •••• | xx(xx.x) |

<sup>\*</sup> Denominator of tabulation is the number of Safety Population

- >Listing for "9.1.2 Summary Table of Concomitant Medication" will be also provided in same format.
- >Row 4 column 3 will be changed to "9.1.2 Summary Table of Concomitant Medication"
- >Row 10 column 3 will be changed to "Subjects with at least one concomitant medication"
- >Sort order;

- 9 Treatments and Medications
- 9.1 Prior and Concomitant Medications
- 9.1.3 Listing of Medications

## Safety population

| Subject<br>Number | Start Date of<br>Study | Start Date [1]/ Do | oute/<br>ose [Units]/<br>equency | Who Drug ATC level 2<br>term/<br>Who Drug ATC level 4<br>term/<br>Preferred Term/<br>Reported Term | Indication |
|---|---|---|---|---|---|
| XX | yyyy-mm-dd | yyyy-mm-dd [88] * OR<br>yyyy-mm-dd [88]<br>yyyy-mm-dd [88] INJ | RAL | vvvvvvvvvv / xxxxxxxxx / yyyyyyyy / 77777777777777 | ADVERSE EVENT (XXXXXXXXXXXX) / PFT |
| xx | yyyy-mm-dd | yyyy-mm-dd [88]<br>yyyy-mm-dd [88] * OT | ГНЕR (SPECIFY) | xxxxxxxxx /<br>yyyyyyyy /<br>77777777777777<br>vvvvvvvvvvv / | OTHERS (XXXXXXXXXXXX) |
| | | yyyy-mm-dd [88] | | xxxxxxxxx /<br>yyyyyyyy /<br>zzzzzzzzzzzzzzz | ADVERSE EVENT (XXXXXXXXXXXX) / |

<sup>\*</sup> New medications starting after the first infusion will be indicated if the medication start date relative to the first study drug infusion is greater than 0

- [1] Study start date =< medication start date: medication start date study start date + 1 Study start date > medication start date: medication start date study start date
- [2] Study start date =< medication end date: medication end date Study start date + 1 Study start date > medication end date: medication end date - Study start date

# >Sort order;

Subject Number, Concomitant Medications Start Date, ATC term, Preferred Term (both alphabetical order)

- 9 Treatments and Medications
- 9.2 Extent of Exposure
  9.2.1 Summary Table of Drug Exposure

| Parameter | |
|------------------------------|-----------|
| Statistics | |
| Treatment duration [week] | |
| N | XX |
| Mean(S.D.) | xx (xx x) |
| Median | XX X |
| Min, Max | xx,xx |
| Number of infusions received | |
| N | XX |
| Mean(S.D.) | xx(xxx) |
| Median | XX X |
| Min, Max | XX, XX |
| Total volume infused [mL] | |
| N | XX |
| Mean(S.D.) | xx(xxx) |
| Median | XX X |
| Min, Max | XX, XX |
| Volume infused per week [mL] | |
| N | XX |
| Mean(S.D.) | |
| Median | XX X |
| Min, Max | XX, XX |
| Infusion duration [minute] | |
| N | XX |
| Mean(S.D.) | xx (xx x) |
| Median | XX X |
| Min, Max | XX,XX |

- 9 Treatments and Medications
- 9.2 Extent of Exposure9.2.2 Summary Table of Infusion Interruptions

| Visit | Number of Infusions | Number of Infusions with Interruption $N$ (%) |
|---|---|---|
| Week 1 | XXX | xx (xx x) |
| Week 2 | XXX | xx (xx x) |
| Week 3 | XXX | xx (xx x) |
| • • • • | •••• | •••• |

<sup>\*</sup> Denominator of tabulation is the number of infusion at the visit

<sup>\*</sup> A subject without infusion at the visit was excluded from analysis

- 9 Treatments and Medications
- 9.2 Extent of Exposure9.2.3 Listing of Exposure Information

# Safety population

| | | Study Drug | | | | | |
|---|---|---|---|---|---|---|---|
| | | Infused/ | Infusion | | Total Volume | | |
| | | Reason for No | Start Date and Time/ | Infusion | Prepared [mL]/ | Infusion Interrupted / | |
| Subject | | Study Drug | Infusion Stop Date and Time | Duration | Total Volume | Explanation for | Reason for less than |
| Number | Visit | Infused | (including saline flush) | [Minutes] | Infused [mL] | Interruption | 100% of IP |
| XX | Week 1 | V | yyyy-mm-ddThh:mm/ | XX X | xxxx/ | N | |
| | | 1 | yyyy-mm-ddThh:mm | | XXXX | 14 | |
| | Week 2 | xxxxxxxxxxxx | yyyy-mm-ddThh:mm/ | XX X | xxxxxxxx/ | xxxxxxxx | |
| | | АЛЛАЛАЛАЛАЛА | yyyy-mm-ddThh:mm | | XXXX | АААААА | |
| XX | Week 1 | V | yyyy-mm-ddThh:mm/ | XX X | xxxxxxxx/ | | xxxxxxx |
| | | 1 | yyyy-mm-ddThh:mm | | XXXX | | ΑΛΛΑΛΑΛ |
| | Week 2 | Y | | | | | |

>Sort order;

Subject Number, Visit

- 9 Treatments and Medications
- 9.3 Treatment Compliance9.3.1 Summary Table of Treatment Compliance

| | N (%) |
|-----------------------------------------------------|-----------|
| Treatment compliance [%] | XX |
| N | xx (xx x) |
| Mean(S.D.) | XX.X |
| Median | XX,XX |
| Min , Max | |
| The number of subjects with treatment compliance >= | xx (xx x) |
| Infusion compliance [%] | |
| N | XX |
| Mean(S.D.) | xx (xx x) |
| Median | XX.X |
| Min, Max | XX,XX |

<sup>\*</sup> Denominator of tabulation is the number of Safety Population

- 9 Treatments and Medications
- 9.3 Treatment Compliance9.3.2 Listing of Treatment Compliance

# Safety population

| Subject | Treatment | | |
|---------|------------|-------|-------------------------|
| Number | Compliance | >=80% | Infusion Compliance [%] |
| XX | XX X | Y | xx x |
| XX | XX X | | |
| XX | XX X | | |

<sup>\*</sup> Treatment compliance = total volume infused / total volume prepared \* 100 [%]

>Sort order; Subject Number

- 10 Exploratory Analysis 10.1 PK Analysis (GTI1401 only) 10.1.1 Summary Table of Alpha1-PI Concentrations

| Alpha1-PI concentrations [mg/dL] | |
|---|---|
| Time Points | |
| Statistics | |
| Immediately before the intravenous infusion | |
| N | XX |
| Mean(S.D.) | xx.x(xxx) |
| %CV | XX.X |
| Median | XX.X |
| Min, Max | XX,XX |
| Geometric mean | XX.X |
| N<br>N | xx |
| Mean(S.D.) | xx.x(xxx) |
| Mean(S.D.)<br>%CV | xx.x (xx x)<br>xx.x |
| Mean(S.D.)<br>%CV<br>Median | xx.x (xx x)<br>xx.x<br>xx.x |
| Mean(S.D.) %CV Median Min , Max | xx.x (xx x)<br>xx.x<br>xx.x<br>xx , xx |
| Mean(S.D.)<br>%CV<br>Median | xx.x (xx x)<br>xx.x<br>xx.x |
| Mean(S.D.) %CV Median Min , Max | xx.x (xx x)<br>xx.x<br>xx.x<br>xx , xx |
| Mean(S.D.) %CV Median Min , Max Geometric mean 15 minutes after completion of the intravenous infusion N | xx.x (xx x)<br>xx.x<br>xx.x<br>xx , xx |
| Mean(S.D.) %CV Median Min , Max Geometric mean 15 minutes after completion of the intravenous infusion | xx.x (xx x) xx.x xx.x xx , xx xx , xx |
| Mean(S.D.) %CV Median Min , Max Geometric mean 15 minutes after completion of the intravenous infusion N Mean(S.D.) %CV | xx.x (xx x) xx.x xx.x xx , xx xx , xx xx.x |
| Mean(S.D.) %CV Median Min , Max Geometric mean 15 minutes after completion of the intravenous infusion N Mean(S.D.) %CV Median | xx.x (xx x) xx.x xx.x xx , xx xx , xx xx.x |
| Mean(S.D.) %CV Median Min , Max Geometric mean 15 minutes after completion of the intravenous infusion N Mean(S.D.) %CV | xx.x (xx x) xx.x xx.x xx , xx xx , xx xx.x |

- 10 Exploratory Analysis
- 10.1 PK Analysis (GTI1401 only)
- 10.1.1 Summary Table of Alpha1-PI Concentrations

### PK population

# Alpha1-PI concentrations [mg/dL]

Time Points

Statistics

| $168 \text{ hours} \pm 1 \text{ day}$ | (7 days after cor | npletion of the intraven | ous infusion) (Week 9) |
|---|---|---|---|

| N | XX |
|----------------|-----------|
| Mean(S.D.) | xx.x(xxx) |
| %CV | XX.X |
| Median | XX.X |
| Min, Max | XX,XX |
| Geometric mean | XX.X |

# >Time points;

- Immediately before the intravenous infusion
- Immediately after the intravenous infusion (after flushing the infusion line with physiological saline) (at 0 hours)
- 15 minutes after completion of the intravenous infusion
- 2 hours after completion of the intravenous infusion
- 4 hours after completion of the intravenous infusion
- 8 hours after completion of the intravenous infusion
- 24  $\pm$  4 hours (1 day after completion of the intravenous infusion)
- 48  $\pm$  4 hours (2 days after completion of the intravenous infusion)
- 120 hours  $\pm$  1 day (5 days after completion of the intravenous infusion)

- 10 Exploratory Analysis 10.1 PK Analysis (GTI1401 only) 10.1.2 Summary Table of Trough (pre-infusion) Levels (Cmin) and mean Cmin

| Cmin [mg/dL] | |
|----------------|-------------|
| Visit | |
| Statistics | |
| Week 1 | |
| N | XX |
| Mean(S.D.) | xx x (xx x) |
| %CV | XX X |
| Median | XX X |
| Min, Max | XX,XX |
| Geometric mean | XX.X |
| Week 7 | |
| N | XX |
| Mean(S.D.) | xx x (xx x) |
| %CV | XX X |
| Median | XX X |
| Min, Max | XX,XX |
| Geometric mean | XX.X |
| Week 8 | |
| N | XX |
| Mean(S.D.) | xx x (xx x) |
| %CV | XX X |
| Median | |
| Min, Max | XX,XX |
| Geometric mean | XX.X |
| Week 9 | |
| N | XX |
| Mean(S.D.) | xx x (xx x) |
| %CV | XX X |
| Median | XX X |
| Min, Max | XX,XX |
| Geometric mean | XX.X |

- 10 Exploratory Analysis 10.1 PK Analysis (GTI1401 only) 10.1.2 Summary Table of Trough (pre-infusion) Levels (Cmin) and mean Cmin

| XX |
|-------------|
| YY |
| YY |
| AA |
| xx x (xx x) |
| XX X |
| XX X |
| XX, XX |
| XX.X |
| xx |

<sup>\*</sup> mean Cmin = Average of Cmin of each patient measured at Week 7, Week 8 and Week 9 (Exclude Week 1)

GTI 1401 10 Exploratory Analysis 10.1 PK Analysis (GTI1401 only) 10.1.3 Figures of Concentration Versus Time Curves of Individual Subjects



GTI 1401

- 10 Exploratory Analysis
  10.1 PK Analysis (GTI1401 only)
  10.1.4 Figures of Concentration Versus Time Curves of All Subjects



- GTI 1401 10 Exploratory Analysis 10.1 PK Analysis (GTI1401 only) 10.1.5 Summary of PK Parameters

| Parameter | Statistics | |
|-------------------------|----------------|-------------|
| AUC0-7days [mg · hr/dL] | N | XX |
| | Mean(S.D.) | xx x (xx x) |
| | %CV | XX X |
| | Median | XX X |
| | Min, Max | XX,XX |
| | Geometric mean | XX X |
| Cmax [mg/dL] | N | XX |
| | Mean(S.D.) | xx x (xx x) |
| | %CV | XX X |
| | Median | XX X |
| | Min, Max | XX,XX |
| | Geometric mean | |
| tmax [hours] | N | XX |
| | Mean(S.D.) | xx x (xx x) |
| | %CV | XX X |
| | Median | XX X |
| | Min, Max | XX,XX |
| t1/2 [hours] | | xx |
| | Mean(S.D.) | xx x (xx x) |
| | %CV | xx x |
| | Median | XX X |
| | Min, Max | XX,XX |
| | Geometric mean | XX X |

GTI 1401 10 Exploratory Analysis 10.1 PK Analysis (GTI1401 only) 10.1.6 Listing of Alpha1-PI Concentrations (Week 8 and 9)

| Subject<br>Number | Actual dos infusion [mL] | se<br>Start/ End Date and<br>Time | Scheduled Plasma Collection Time | Exclude<br>from<br>PK<br>Analysis | Nominal<br>Time<br>Point<br>[hr] | Actual Plasma Collection<br>Date / Time | Elapsed<br>Times from<br>the Start of<br>the Study<br>Drug<br>Infusion [hr] | Value of Alpha-<br>PI<br>Concentrations<br>[mg/dL] |
|---|---|---|---|---|---|---|---|---|
| xxxx | xx | yyyy-mm-ddThh mm/<br>yyyy-mm-ddThh mm | IMMEDIATELY BEFORE THE INTRAVENOUS INFUSION IMMEDIATELY AFTER THE INTRAVENOUS | | 0 | yyyy-mm-ddThh mm | xx | xxx xx |
| | | | INFUSION | | 0.25 | yyyy-mm-ddThh mm | XX | xxx xx |
| | | | 15 MINUTES AFTER COMPLETION OF THE INTRAVENOUS INFUSION | Y | 0.5 | yyyy-mm-ddThh mm | xx | xxx xx |
| | | | 2 HOURS AFTER COMPLETION OF THE INTRAVENOUS INFUSION | | 2.25 | yyyy-mm-ddThh mm | xx | xxx xx |
| | | | 4 HOURS AFTER COMPLETION OF THE INTRAVENOUS INFUSION | | 4.25 | yyyy-mm-ddThh mm | xx | BLQ<br>xxx xx |
| xxxx | xx | yyyy-mm-ddThh mm/<br>yyyy-mm-ddThh mm | IMMEDIATELY BEFORE THE INTRAVENOUS INFUSION | | 0 | yyyy-mm-ddThh mm | xx | xxx xx |
| | | | IMMEDIATELY AFTER THE INTRAVENOUS INFUSION | | 0.25 | yyyy-mm-ddThh mm | xx | xxx xx |
| | | | 15 MINUTES AFTER COMPLETION OF THE INTRAVENOUS INFUSION | | 0.5 | yyyy-mm-ddThh mm | xx | xxx xx |
| | | | 2 HOURS AFTER COMPLETION OF THE INTRAVENOUS INFUSION | | 2.25 | yyyy-mm-ddThh mm | XX | xxx xx |

<sup>\*</sup> BLQ: Below limit of quantification
10 Exploratory Analysis 10.1 PK Analysis (GTI1401 only) 10.1.6 Listing of Alpha1-PI Concentrations (Week 8 and 9)

PK population

| | | | | | | | Elapsed | |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | Times from | |
| | | | | Exclude | Nominal | | the Start of | Value of Alpha- |
| | Actual dose | ; | | from | Time | | the Study | PI |
| Subject | infusion | Start/ End Date and | | PK | Point | Actual Plasma Collection | Drug | Concentrations |
| Number | [mL] | Time | Scheduled Plasma Collection Time | Analysis | [hr] | Date / Time | Infusion [hr] | [mg/dL] |

>Sort order;

Subject Number, Nominal Time Point [hr]

10 Exploratory Analysis 10.1 PK Analysis (GTI1401 only) 10.1.7 Listing of Alpha1-PI Concentrations

# PK population

| | Scheduled Plasma | Exclude from | Actual Plasma Collection Date / | Value of<br>Alpha-PI<br>Concentrations |
|---|---|---|---|---|
| Subject Number | Collection Visit | PK Analysis | Time | [mg/dL] |
| XXXX | SCREENING | Y | yyyy-mm-ddThh:mm | XXX.XX |
| | Week 1 | | yyyy-mm-ddThh:mm | XXX.XX |
| | Week 7 | | yyyy-mm-ddThh:mm | XXX.XX |
| ••••• | | • | | |
| XXXX | SCREENING | Y | yyyy-mm-ddThh:mm | XXX.XX |
| | Week 1 | | yyyy-mm-ddThh:mm | XXX.XX |
| | Week 7 | | yyyy-mm-ddThh:mm | xxx.xx |

<sup>\*</sup> BLQ: Below limit of quantification

# >Sort order;

Subject Number, Scheduled Plasma Collection Visit, Actual Plasma Collection Date / Time

10 Exploratory Analysis

10.1 PK Analysis (GTI1401 only) 10.1.8 Listing of Trough (pre-infusion) levels (Cmin) and mean Cmin

# PK population

| Subject Number | Visit | Trough Level Cmin [mg/dL] |
|----------------|-------------|---------------------------|
| XXXX | Week 1 | XXX |
| | Week 7 | XXX |
| | Week 8 | XXX |
| | Week 9 | XXX |
| | Mean Cmin * | XXX |
| XXXX | Week 1 | XXX |
| | Week 7 | XXX |
| | Week 8 | XXX |
| | Week 9 | XXX |
| | Mean Cmin * | XXX |

<sup>\*</sup> mean Cmin = Average of Cmin of each patient measured at Week 7, Week 8 and Week 9 (Exclude Week 1)

>Sort order;

Subject Number, Visit (Mean Cmean appear at last record within subject)

- GTI 1401 10 Exploratory Analysis 10.1 PK Analysis (GTI1401 only) 10.1.9 Listing of PK Parameters

# PK population

| Subject Number | AUC0-7days [mg · hr/dL] | Cmax [mg/dL] | tmax [hours] | t1/2 [hours] | Cmin [mg/dL] |
|---|---|---|---|---|---|
| XXXX | XXXX | XXXX | XXX | XXX | XXX |
| XXXX | XXXX | XXXX | XXX | XXX | XXX |
| XXXX | XXXX | XXXX | XXX | XXX | XXX |

>Sort order; Subject Number

- 10 Exploratory Analysis 10.2 Lung Density Analysis (GTI1401 only) 10.2.1 Summary Table of Lung Density

# Safety population

| Parameter [unit] | Location | Statistics | |
|------------------------|-------------------------|------------|-----------|
| Hu value 15 percentile | LUNG | N | XX |
| 10/1.1 | | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | xx,xx |
| | LUNG, LEFT | N | XX |
| | | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | xx, $xx$ |
| | LUNG, LEFT LOWER LOBE | N | XX |
| | | Mean(S.D.) | xx(xxx) |
| | | Median | XX X |
| | | Min, Max | XX, XX |
| | LUNG, LEFT UPPER LOBE | N | XX |
| | | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | XX, XX |
| | LUNG, RIGHT | N | XX |
| | | Mean(S.D.) | xx(xxx) |
| | | Median | XX X |
| | | Min, Max | XX, XX |
| | LUNG, RIGHT LOWER LOBE | N | XX |
| | | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | XX,XX |
| | LUNG, RIGHT MIDDLE LOBE | N | xx |
| | | Mean(S.D.) | xx(xxx) |
| | | Median | XX X |

- 10 Exploratory Analysis 10.2 Lung Density Analysis (GTI1401 only) 10.2.1 Summary Table of Lung Density

# Safety population

| Parameter [unit] | Location | Statistics | |
|------------------|-------------------------|------------|-----------|
| | | Min, Max | XX, XX |
| | LUNG, RIGHT UPPER LOBE | N | XX |
| | | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | XX, XX |
| | LUNG, THIRDS LEFT LOWER | N | XX |
| | | Mean(S.D.) | xx(xxx) |
| | | Median | xx x |
| | | Min, Max | XX, XX |
| | LUNG, THIRDS LEFT MIDDL | E N | XX |
| | , | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | XX, XX |
| | LUNG, THIRDS LEFT UPPER | N | XX |
| | | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | xx,xx |
| | LUNG, THIRDS RIGHT LOWE | ERN | XX |
| | | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | XX, XX |
| | LUNG, THIRDS RIGHT MIDD | L' N | xx |
| | | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | xx,xx |
| | LUNG, THIRDS RIGHT UPPE | RN | XX |
| | | Mean(S.D.) | xx (xx x) |

10 Exploratory Analysis

10.2 Lung Density Analysis (GTI1401 only)

10.2.1 Summary Table of Lung Density

### Safety population

| Parameter [unit] | Location | Statistics | |
|------------------------|----------|------------|-----------|
| • | | Median | xx x |
| | | Min, Max | XX, XX |
| Mean [hounsfield unit] | LUNG | N | XX |
| | | Mean(S.D.) | xx (xx x) |
| | | Median | XX X |
| | | Min, Max | XX,XX |
| | •••• | •••• | •••• |

All location for following parameters will be displayed after Air Volume in cm3;

Mean [g/L]

Standard deviation [g/L]

Percent below -856 hu [%]

Percent below -910 hu [%]

Percent below -950 hu [%]

Total volume in cm3 [mL]

Air volume in cm3 [mL]

Tissue volume in cm3 [mL]

GTI 1401 10 Exploratory Analysis 10.2 Lung Density Analysis (GTI1401 only) 10.2.2 Listing of Lung Density

| Subject Number | Location | Hu Value 15 Percentile [g/L] | Mean [g/L] | Standard<br>deviation<br>[g/L] | Percent<br>below -856<br>hu [%] | Percent<br>below -910<br>hu [%] | Percent<br>below -950<br>hu [%] | Total volume in cm3 [mL] | Air volume in cm3 [mL] | Tissue volume in cm3 [mL] |
|---|---|---|---|---|---|---|---|---|---|---|
| XXXX | LUNG | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| | LUNG, LEFT | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| | LUNG, LEFT LOWER LOBE | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| | LUNG, LEFT UPPER LOBE | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| | LUNG, RIGHT | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | xx x |
| | LUNG, RIGHT LOWER LOBE | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | xx x |
| | LUNG, RIGHT MIDDLE LOBE | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| | LUNG, RIGHT UPPER LOBE | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | xx x |
| | LUNG, THIRDS LEFT LOWER | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| | LUNG, THIRDS LEFT MIDDLE | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | xx x |
| | LUNG, THIRDS LEFT UPPER | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| | LUNG, THIRDS RIGHT LOWER | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| | LUNG, THIRDS RIGHT MIDDLE | XX X | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| | LUNG, THIRDS RIGHT UPPER | xx x | XX X | XX.X | XX X | XX X | XX X | XX X | XX.X | XX X |
| xxxx | LUNG | xx x | XX X | XX.X | XX X | xx x | XX X | XX X | xx.x | XX X |

>Sort order; Subject Number, Location

GTI 1401 11 Safety Analysis 11.1 Adverse Events 11.1.1 Overview of AEs

# Safety population

| | N=88 |
|---|---|
| | n (%) |
| The number of subjects with at least one AE | xx (xx x) |
| The number of AE | XX |
| The number of subject with at least one ADR | xx (xx x) |
| The number of events with ADR | XX |
| The number of subject with at least one AE with fatal outcome | xx (xx x) |
| The number of AE with fatal outcome | XX |
| The number of subject with at least one SAE | xx (xx x) |
| The number of SAE | XX |
| The number of subject with at least one AE leading to premature discontinuation from the study | xx (xx x) |
| The number of AE leading to premature discontinuation from the study | xx |
| The number of subject with at least one event of Special Interest | xx (xx x) |
| The number of event of Special Interest | XX |

<sup>\*</sup> Denominator of tabulation is the number of Safety population

- 11 Safety Analysis
- 11.1 Adverse Events
- 11.1.2 Summary Table of AEs

#### Safety population

| | N=88 |
|---------------------------------------------|-----------|
| | n (%) |
| The number of AE | XX |
| The number of subjects with at least one AE | xx (xx x) |
| SOC1 | xx (xx x) |
| PT1 | xx(xxx) |
| SOC2 | xx(xxx) |
| PT2 | xx(xxx) |

<sup>\*</sup> Denominator of tabulation is the number of Safety population

>Table for "11.1.3 Summary Table of ADRs" will be also provided in same layout.

>Row 4 column 3 will be changed to "11.1.3 Summary Table of ADRs"

>Row 10 column 3 will be changed to "The number of ADR"

>Row 12 column 3 will be changed to "The number of subjects with at least one ADR".

>Sort order;

SOC name, PT name (Both alphabetical order)

- 11 Safety Analysis
- 11.1 Adverse Events
- 11.1.4 Summary Table of AEs by Causality

### Safety population

| | N=88 | | | | |
|---|---|---|---|---|---|
| | Definite | Probable | Possible | Doubtful/Unlikel | Unrelated |
| | n (%) | n (%) | n (%) | у | n (%) |
| The number of AE | xx/108 | xx/108 | xx/108 | xx/108 (xx x) | xx/108 |
| The number of subjects with at least one AE | xx (xx.x) | xx (xx.x) | xx (xx x) | xx (xx x) | xx (xx.x) |
| SOC1 | xx (xx.x) | xx (xx.x) | xx (xx x) | xx (xx x) | xx (xx.x) |
| PT1 | xx (xx.x) | xx (xx.x) | xx (xx x) | xx(xxx) | xx (xx.x) |
| SOC2 | xx (xx.x) | xx (xx.x) | xx (xx x) | xx(xxx) | xx (xx.x) |
| PT2 | xx (xx.x) | xx (xx.x) | xx (xx x) | xx(xxx) | xx (xx.x) |

>Sort order;

SOC name, PT name (Both alphabetical order)

<sup>\*</sup> Denominator of tabulation is the number of Safety population
\* If a subject experiences the same adverse event with more than one relationship to study drug, the stronger causal relationship to study drug will be counted only once in the total of those experiencing adverse events in that particular

- 11 Safety Analysis
- 11.1 Adverse Events
- 11.1.5 Summary Table of AEs by Severity

#### Safety population

| | N=88 | | |
|---|---|---|---|
| | Mild | Moderate | Severe |
| | n (%) | n (%) | n (%) |
| The number of AE | xx/108 (xx.x) | xx/108 (xx.x) | xx/108 (xx.x) |
| The number of subjects with at least one AE | xx (xx x) | xx(xxx) | xx (xx x) |
| SOC1 | xx (xx x) | xx (xx x) | xx (xx x) |
| PT1 | xx (xx x) | xx (xx x) | xx (xx x) |
| SOC2 | | | |
| PT2 | ••• | • • • | ••• |

<sup>\*</sup> Denominator of tabulation is the number of Safety population

>Listing for "11.1.6 Summary Table of ADRs by Severity" will be also provided in same layout.

- >Row 4 column 3 will be changed to "11.1.6 Summary Table of ADRs by Severity"
- >Row 10 column 3 will be changed to "The number of ADR"
- >Row 12 column 3 will be changed to "The number of subjects with at least one ADR".

>Sort order;

SOC name, PT name (Both alphabetical order)

<sup>\*</sup> If a subject experiences the same adverse event at more than one severity, the most severe rating to study drug will be counted only once in the total of those experiencing adverse events in that particular system organ class / preferred term.

GTI 1401 11 Safety Analysis

11.1 Adverse Events

11.1.7 Listing of AEs

Safety population

| Subject | Start / End Date and Time | Relative | MedDRA System Organ<br>Class/<br>Preferred Term/ | Pattern/<br>Seriousness / Severity /<br>Action Taken with | Causality to<br>Study Drug / | | | Concomitant Medication/ |
|---|---|---|---|---|---|---|---|---|
| Number | of Events | days * | Verbatim Term | Study Drug | Outcome | (a) | (b) | Other Action |
| XXXX | yyyy-mm-ddThh:mm/ | X | xxxx/ | INTERMITTENT/ | DOUBTFUL/UN | Y | N | N/ |
| | yyyy-mm-ddThh:mm | | уууу/ | N / | LIKELY/ | | | N |
| | | | ZZZZ | MILD / | RECOVERING/ | | | |
| | | | | DRUG WITHDRAWN | RESOLVING | | | |
| xxxx | yyyy-mm-ddThh:mm/ | X | | CONTINUOUS/ | DEFINITE / | Y | Y | N/ |
| | yyyy-mm-ddThh:mm | | | N/ | RECOVERED / | | | N |
| | | | | MILD / | RESOLVED | | | |
| | | | | MODERATE | WITH | | | |
| xxxx | yyyy-mm-ddThh:mm/ | X | xxxx/yyyy/zzzz<br>xxxx/ | CONTINUOUS | DEFINITE / | | N | Y (xxxxx)/ |
| | yyyy-mm-ddThh:mm | | уууу/ | N/ | RECOVERED / | | | Y (xxxxx) |
| | | | ZZZZ | MILD / | RESOLVED | | | |
| | | | | MODERATE | WITH | | | |
| | ••• | | ••• | ••• | | | | |

<sup>\*</sup> Study start date =< Onset date of event: Onset date of event - Study start date +

Study start date > Onset date of event: Onset date of event - Study start date \* (a)TEAE  $\,/\,$  (b)Did the subject withdraw from the study?

>Listing for "11.1.11 Listing of AEs leading to Premature Discontinuation from the Study" will be also provided in same layout. >Row 4 column 3 will be changed to "11.1.11Listing of AEs leading to Premature Discontinuation from the Study"

>Sort order;

<sup>1,</sup> 

- 11 Safety Analysis
- 11.1 Adverse Events
- 11.1.8 Listing of Death

Safety population

| Subject<br>Number | Start / End Date of<br>Events | Relative days <sup>[1]</sup> | Date of Death [Relative days] <sup>[2]</sup> | MedDRA System<br>Organ Class/<br>Preferred Term/<br>Verbatim Term | Pattern/<br>Seriousness / Severity /<br>Action Taken with<br>Study Drug | Causality to<br>Study Drug /<br>Outcome | (a) | (b) | Concomitant Medication/ Other Action/ Cause of Death |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | , , | DOUBTFUL/UN | (a) | ( ) | |
| XXXX | yyyy-mm-ddThh:mm | X | yyyy-mm-dd | xxxx/ | INTERMITTENT/ | | Y | N | N/ |
| | / | | [x] | уууу/ | N / | LIKELY/ | | | N/ |
| | yyyy-mm-ddThh:mm | | | ZZZZ | MILD / | RECOVERING/ | | | xxxxxxxxxxxxxxxxxxxxxxx |
| | | | | | DRUG WITHDRAWN | RESOLVING | | | xxxxxxxxx |
| xxxx | yyyy-mm-ddThh:mm | X | | xxxx/ | CONTINUOUS/ | DEFINITE / | Y | Y | N/ |
| | / | | | yyyy/ | N/ | RECOVERED / | | | N/ |
| | yyyy-mm-ddThh:mm | | | ZZZZ | MILD / | RESOLVED | | | xxxxxxxxxx |
| | | | | | MODERATE | WITH | | | |
| | 1.1771.1 | | | , | CONTRIBUTION | CEULIEL VE | | | <b>T</b> |
| XXXX | yyyy-mm-ddThh:mm | X | | XXXX/ | CONTINUOUS | DEFINITE / | | N | Y (xxxxx)/ |
| | / | | | yyyy/ | N/ | RECOVERED / | | | Y (xxxxx)/ |
| | yyyy-mm-ddThh:mm | | | ZZZZ | MILD / | RESOLVED | | | xxxxxxxxxxxxxxxxxx |
| | | | | | MODERATE | WITH | | | |
| | ••• | | | | ••• | | | | |

<sup>\* [1]</sup> Study start date =< Onset date of event: Onset date of event - Study start date + 1, Study start date > Onset date of event: Onset date of event - Study start date

# >Sort order;

Subject Number, Start Date of Events, Start Time of Events Outcome of AEs is death will be listed.

<sup>\* [2]</sup>Date of death - study start date + 1
\* (a)TEAE / (b)Did the subject withdraw from the study?

- 11 Safety Analysis
- 11.1 Adverse Events
- 11.1.9 Listing of SAE

Safety population

| | | | MedDRA System Organ<br>Class/ | Pattern/<br>Seriousness / Severity | Causality to | | | Concomitant | Reason |
|---|---|---|---|---|---|---|---|---|---|
| Subject | Start / End Date and Time | Relative | Preferred Term/ | Action Taken with | Study Drug / | | | Medication/ | Seriousness / |
| Number | of Events | days * | Verbatim Term | Study Drug | Outcome | (a) | (b) | Other Action | Detail |
| xxxx | yyyy-mm-ddThh:mm/ | X | xxxx/ | INTERMITTENT/ | DOUBTFUL/UN | Y | N | N/ | RESULT IN DEATH / |
| | yyyy-mm-ddThh:mm | | уууу/ | N / SEVERE | LIKELY/ | | | N | xxxxxxxxxxxxxxx |
| | | | ZZZZ | DRUG WITHDRAWN | RECOVERING/ | | | | XX |
| | | | | | RESOLVING | | | | |
| xxxx | yyyy-mm-ddThh:mm /<br>yyyy-mm-ddThh:mm | X | xxxx/yyyy/zzzz | CONTINUOUS/<br>N/ SEVERE | DEFINITE /<br>RECOVERED / | Y | Y | N/<br>N | LIFE-THREATENING |
| | | | | MODERATE | RESOLVED | | | | |
| | | | | | WITH | | | | |
| xxxx | yyyy-mm-ddThh:mm /<br>yyyy-mm-ddThh:mm | x | xxxx/<br>yyyy/<br>zzzz | CONTINUOUS<br>N/ SEVERE<br>MODERATE | DEFINITE / RECOVERED / RESOLVED WITH | | N | Y (xxxxx)/<br>Y (xxxxx) | IMPORTANT MEDICAL EVENT (xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| • • • | ••• | | ••• | ••• | • • • | | | | |

<sup>\*</sup> Study start date =< Onset date of event: Onset date of event - Study start date +

Study start date > Onset date of event: Onset date of event - Study start date \* (a)TEAE / (b)Did the subject withdraw from the study?

>Sort order;

Subject Number, Start Date of Events, Start Time of Events

- 11 Safety Analysis
- 11.1 Adverse Events
- 11.1.11 Listing of Non-Serious COPD Exacerbation

Safety population

| Subject | Start / End Date and Time of | Relative | Pattern/ | Action Taken with | Causality to Study | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Events | days* | Severity | Study Drug | Drug | Outcome | (a) | (b) | (c) | (d) | (e) | (f) |
| XXXX | yyyy-mm-ddThh:mm / | X | INTERMITTENT/ | | | RECOVERING/ | | | | | | |
| | yyyy-mm-ddThh:mm | | MILD | DRUG WITHDRAWN | | RESOLVING<br>RECOVERED / | Y | N | N | N | N | N |
| | yyyy-mm-ddThh:mm/ | X | CONTINUOUS/ | DOSE NOT | | RESOLVED WITH | | | | Y/Y/ | | |
| XXX | yyyy-mm-ddThh:mm | | MODERATE | CHANGED | DEFINITE | SEQUELAE<br>RECOVERED / | Y | Y | Y | CLEAR | Y | N |
| | yyyy-mm-ddThh:mm/ | X | CONTINUOUS/ | DOSE NOT | | RESOLVED WITH | | | | | | |
| XXXX | yyyy-mm-ddThh:mm | | MODERATE | CHANGED | DEFINITE | SEQUELAE | Y | N | N | N | N | N |
| | ••• | | | | | | | | | | | |

<sup>\*</sup> Study start date =< Onset date of event: Onset date of event - Study start date + 1, Study start date > Onset date of event: Onset date of event - Study start date

>Sort order;

Subject Number, Start Date of Events, Start Time of Events

<sup>\* (</sup>a)Did the subject withdraw from the study as a result of this event? / (b)Did the subject experience increased dyspnea? / (c)Did the subject experience increased cough? / (d)Did the subject expectorate sputum?/ more than usual?/ The color / (e)Did the subject increase their usual treatment? / (f)Did the subject take antibiotics or oral steroids?

- 11 Safety Analysis
- 11.2 Laboratory tests
  11.2.1 Summary Table of Laboratory Test

# Safety population Albumin [g/L]

| Visit | | |
|------------|----------------|----------------------|
| Statistics | Original Value | Change from Baseline |
| Baseline | | |
| N | xx x | - |
| Mean(S.D.) | xx.x (xx x.) | - |
| Median | xx x | - |
| Min, Max | XX X , XX.X | - |
| Week 5 | | |
| N | xx x | XX X |
| Mean(S.D.) | xx.x (xx x.) | xx x (xx.x.) |
| Median | xx x | XX X |
| Min, Max | XX X , XX.X | xx x , xx x |
| Week 9 | | |
| N | xx x | XX X |
| Mean(S.D.) | xx.x (xx x.) | xx x (xx.x.) |
| Median | xx x | XX X |
| Min, Max | xx x , xx.x | XX X , XX X |

>All chemistry and hematology laboratory parameter will be summarized in same layout.

>Row 7 column 3 will be changed by the laboratory parameter.

- 11 Safety Analysis
- 11.2 Laboratory tests
  11.2.2 Summary Shift Table of Laboratory Test (Low, Normal and High)

# Safety population

### Albumin

| | | | Baseline | | |
|---------|-----|--------|----------|---------|-------|
| | Low | Normal | High | Missing | Total |
| Week 5 | | | | | |
| Low | XX | XX | XX | XX | XX |
| Normal | XX | XX | XX | XX | XX |
| High | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX |
| Total | xx | XX | XX | XX | XX |
| Week 9 | | | | | |
| Low | XX | XX | XX | XX | XX |
| Normal | XX | XX | XX | XX | XX |
| High | XX | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX | XX |
| Total | XX | XX | XX | XX | XX |

>All chemistry and hematology laboratory parameter will be summarized in same layout.

>Row 7 column 3 will be changed by the laboratory parameter.

- 11 Safety Analysis
- 11.2 Laboratory tests
- 11.2.3 Summary Shift Table of Laboratory Test (Normal and Abnormal)

# Safety population

рΗ

| | | Bas | eline | |
|----------|--------|----------|---------|-------|
| | Normal | Abnormal | Missing | Total |
| Week 5 | | | | |
| Normal | XX | XX | XX | XX |
| Abnormal | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX |
| Total | XX | XX | XX | XX |
| Week 9 | | | | |
| Normal | XX | XX | XX | xx |
| Abnormal | XX | XX | XX | XX |
| Missing | XX | XX | XX | XX |
| Total | XX | XX | XX | XX |

>All urine parameter will be summarized in same layout.

>Row 7 column 3 will be changed by the laboratory

- 11 Safety Analysis
- 11.2 Laboratory tests
  11.2.3 Listing of Laboratory Parameters

Safety population

| Subject<br>Number | Parameter | Visit | Baseline | Date of Sample Collection | Standard Value | Change from Baseline | Normal Range |
|---|---|---|---|---|---|---|---|
| XXXX | Albumin [g/L] | Week 1 | Y | yyyy-mm-dd | xx/H | | xx< <xx< td=""></xx<> |
| xxxx | Alkaline Phosphatase | Week 5<br>Week 9<br>Week 1<br>Week 5<br>Week 9 | Y | yyyy-mm-dd<br>yyyy-mm-dd<br>yyyy-mm-dd<br>yyyy-mm-dd<br>yyyy-mm-dd | xx<br>xx/L<br>xx<br>xx<br>xx | xx<br>xx<br>xx<br>xx | xx< <xx<br>xx&lt; <xx<br>xx&lt; <xx<br>xx&lt; <xx< td=""></xx<></xx<br></xx<br></xx<br> |

<sup>\* &#</sup>x27;H' / 'L' indicates value is higher / lower than normal range respectively.

>Sort order;

Subject Number, Parameter (alphabetical order), Date of Sample Collection

11 Safety Analysis
11.3 Vital Signs
11.3.1 Summary Table of Vital Signs

Safety population

Pulse rate [BEATS/MIN]
Parameter

| Parameter | | |
|---|---|---|
| Visit | | |
| Statistics | Original Value | Change from Baseline |
| Week 1 IMMEDIATELY PRIOR TO START OF INFUSION (Baseline | ) | |
| N | XX X | - |
| Mean(S.D.) | xx x (xx x.) | - |
| Median | XX X | - |
| Min, Max | XX X , XX.X | - |
| Week 1 IMMEDIATELY AFTER COMPLETION OF INFUSION | | |
| N | XX X | XX X |
| Mean(S.D.) | xx x (xx x.) | xx x (xx x.) |
| Median | XX X | xx x |
| Min , Max | xx x , xx.x | xx x , xx x |
| Week 2 IMMEDIATELY PRIOR TO START OF INFUSION | | |
| N | XX X | xx x |
| Mean(S.D.) | xx x (xx x.) | xx x (xx x.) |
| Median | XX X | XX X |
| Min, Max | xx x , xx.x | xx x, xx x |
| Week 2 IMMEDIATELY AFTER COMPLETION OF INFUSION | | |
| N | XX X | xx x |
| Mean(S.D.) | | xx x (xx x.) |
| Median | XX X | xx x |
| Min, Max | XX X, XX.X | xx x , xx x |
| • • • | | |
| Week 9 IMMEDIATELY AFTER COMPLETION OF INFUSION | | |
| N | XX X | xx x |
| Mean(S.D.) | xx x (xx x.) | xx x (xx x.) |
| Median | XX X | XX X |
| Min, Max | XX X , XX.X | xx x , xx x |

11 Safety Analysis

11.3 Vital Signs

11.3.1 Summary Table of Vital Signs

Safety population

Pulse rate [BEATS/MIN]
Parameter

Visit

Original Value Change from Baseline Statistics

>Following vital sign parameter will be summarized in same layout.

"Systolic blood pressure [mmHg]"

"Diastolic blood pressure [mmHg]"

"Body Temperature [C]"

"Respiratory rate [breaths per minute]"

>Row 7 column 3 will be changed by vital sign parameter to following;

"Systolic bloodp pressure [mmHg]"

"Diastolic blood pressure [mmHg]"

"Body temperature [C]"

"Respiratory rate [breaths per minute]"

GTI 1401 11 Safety Analysis 11.3 Vital Signs 11.3.2 Listing of Vital Signs

# Safety population

| Subject | | | | | | from |
|---|---|---|---|---|---|---|
| Number | Parameter | Visit | Baseline | Date / time of Sample Collection | Original Value | baseline |
| XXXX | Pulse rate[BEATS/MIN] | Week 1 IMMEDIATELY PRIOR TO START OF | Y | yyyy-mm-ddThh mm | 100 | - |
| | | Week 1 IMMEDIATELY AFTER COMPLETION OF | | yyyy-mm-ddThh mm | 105 | 121 |
| | | INFUSION | | | | |
| | | Week 2 IMMEDIATELY PRIOR TO START OF | | | | |
| | | Week 2 IMMEDIATELY AFTER COMPLETION OF | | yyyy-mm-ddThh mm | 98 | 125 |
| | | INFUSION | | | | |
| | | ••••• | | ••••• | • • • • • • | • • • • • |
| | Systolic blood pressure [mmHg] | Week 1 IMMEDIATELY PRIOR TO START OF | Y | | | |
| | Diastolic blood pressure [mmHg] | Week 1 IMMEDIATELY PRIOR TO START OF | Y | | | |
| | Body temperature [C] | Week 1 IMMEDIATELY PRIOR TO START OF | Y | yyyy-mm-ddThh mm | XX | - |
| | Respiratory rate [breaths per minute] | Week 1 IMMEDIATELY PRIOR TO START OF | Y | yyyy-mm-ddThh mm | XX | - |
| | | ••••• | | ••••• | ••••• | • • • • • |
| XXXX | Pulse rate[BEATS/MIN] | Week 1 IMMEDIATELY PRIOR TO START OF | Y | yyyy-mm-ddThh mm | XX | - |



- GTI 1401 11 Safety Analysis 11.4 Electrocardiogram 11.4.1 Summary Table of Electrocardiogram

| | | N=88<br>Baseline | | | |
|---|---|---|---|---|---|
| Electrocardio | gram | Normal | Abnormal | Missing | Total |
| Week 9 | Normal | XX | XX | XX | XX |
| | Abnormal | XX | XX | XX | XX |
| | Missing | XX | XX | XX | XX |
| | Total | XX | XX | XX | XX |

> Analysis visit for 1401-OLE;

Baseline

Ext Week 26

Ext Week 52

- GTI 1401 11 Safety Analysis 11.4 Electrocardiogram 11.4.2 Listing of Electrocardiogram

| Subject | | | Electrocardiogram | |
|---|---|---|---|---|
| Number | Visit | Baseline | Performed | Value |
| xxxx | Week 1<br>Week 9 | Y | yyyy-mm-dd<br>yyyy-mm-dd | NORMAL<br>NORMAL |
| xxxx | Week 1<br>Week 9 | Y | yyyy-mm-dd<br>yyyy-mm-dd | ABNORMAL<br>ABNORMAL |

>Sort order; Subject Number, Visit

- GTI 1401 11 Safety Analysis 11.5 Urine Cotinine Tests 11.5.1 Summary Table of Urine Cotinine Test

| | | | N=8 | | |
|---------------------|----------|----------|----------|---------|-------|
| | | Baseline | | | |
| Urine Cotinine Test | | Negative | Positive | Missing | Total |
| Week 5 | Negative | XX | XX | XX | XX |
| | Positive | XX | XX | XX | XX |
| | Total | xx | XX | XX | XX |
| Week 9 | Negative | xx | XX | XX | XX |
| | Positive | XX | XX | XX | XX |
| | Total | XX | XX | XX | XX |

> Analysis visit for 1401-OLE; Baseline Ext Week 26

Ext Week 52

- GTI 1401 11 Safety Analysis 11.5 Urine Cotinine Test 11.5.2 Listing of Urine Cotinine Test

| Subject | | | Date of Sample | |
|---------|---------|----------|----------------|----------|
| Number | Visit | Baseline | Collection | Value |
| XXXX | SCREENI | NG Y | yyyy-mm-dd | NEGATIVE |
| | Week 5 | | yyyy-mm-dd | NEGATIVE |
| | Week 9 | | yyyy-mm-dd | NEGATIVE |
| xxxx | SCREENI | NG Y | yyyy-mm-dd | POSITIVE |
| | Week 5 | | yyyy-mm-dd | POSITIVE |
| | Week 9 | | yyyy-mm-dd | POSITIVE |
| | ••• | ••• | ••• | ••• |

>Sort order; Subject Number, Visit

- 11 Safety Analysis
- 11.6 Pulmonary Function Tests
  11.6.1 Summary Table of Pulmonary Function Tests (FEV1 and FVC)

### Safety population

### PRE-BRONCHODILATOR

| Best FEV [L | | V [L] | Best FVC [L] | | FEV1 pre | dicted [%] |
|---|---|---|---|---|---|---|
| | | Change from | | Change from | | Change from |
| Visit | Original Value | Baseline | Original Value | Baseline | Original Value | Baseline |
| SCREENING | | | | | | |
| N | xx x | - | XX X | - | XX X | - |
| Mean(S.D.) | xx x (xx x) | - | xx x (xx.x) | - | xx.x (xx.x) | - |
| Median | XX X | - | XX X | - | XX.X | - |
| Min, Max | xx x , xx x | - | xx.x , xx x | - | xx x , xx x | - |
| Week 5 | | | | | | |
| N | XX X | XX.X | xx x | xx x | XX X | xx.x |
| Mean(S.D.) | xx x (xx x) | xx.x (xx.x) | xx x (xx.x) | xx x (xx x) | xx.x (xx.x) | xx.x(xxx) |
| Median | xx x | XX.X | XX X | XX X | XX X | xx.x |
| Min, Max | xx x , xx x | xx x , xx x | XX.X , XX X | xx x , xx x | xx x , xx x | XX X , XX X |
| Week 9 | | | | | | |
| N | | XX.X | xx x | xx x | XX X | xx.x |
| Mean(S.D.) | xx x (xx x) | xx.x (xx.x) | xx x (xx.x) | xx x (xx x) | xx.x (xx.x) | xx.x (xx x) |
| Median | xx x | XX.X | XX X | XX X | XX X | xx.x |
| Min, Max | xx x , xx x | xx x , xx x | xx.x, xx x | xx x , xx x | xx x, xx x | xx x , xx x |

>Value for "POST-BRONCHODILATOR" will be summarized after "PRE-BRONCHODILATOR"

>Row 7 and column 3 will be change to "POST-BRONCHODILATOR"

>Analysis visit for 1401-OLE;

-SCREENING (Baseline), Ext Week 26, Ext Week 52

- 11 Safety Analysis
- 11.6 Pulmonary Function Tests
  11.6.2 Summary Table of Pulmonary Function Tests (FEV1 % Predicted)

### Safety population

### PRE-BRONCHODILATOR

| FEV1 % predicted Visit | N=88 |
|------------------------|-----------|
| Statistics | n |
| SCREENING | |
| 0=< < 30 | - |
| 30=< < 70 | xx (xx.x) |
| 70=<<100 | - |
| Missing | - |
| Total | - |
| Week 5 | |
| 0=< < 30 | xx (xx.x) |
| 30=< < 70 | xx (xx.x) |
| 70=<<100 | xx (xx.x) |
| Missing | xx (xx.x) |
| Total | xx (xx.x) |
| Week 9 | |
| 0=< < 30 | xx (xx.x) |
| 30=< < 70 | xx (xx.x) |
| 70=<<100 | xx (xx.x) |
| Missing | xx (xx.x) |
| Total | xx (xx.x) |

>Value for "POST-BRONCHODILATOR" will be summarized after "PRE-BRONCHODILATOR"

>Row 7 and column 3 will be change to "POST-BRONCHODILATOR"

>Analysis visit for 1401-OLE;

- GTI 1401 11 Safety Analysis 11.6 Pulmonary Function Tests 11.6.3 Listing of Pulmonary Function Tests

| | | | | | | Change |
|---|---|---|---|---|---|---|
| Subject | | | | Date / Time of Sample | | from |
| Number | Parameter | Visit | Baseline | Collection | Original Value | Baseline |
| XXXX | Best FEV1 [L] | SCREENING (PRE-BRONCHODILATOR) | Y | yyyy-mm-ddThh:mm | XX | - |
| | | Week 5 (PRE-BRONCHODILATOR) | | yyyy-mm-ddThh:mm | XX | XX |
| | | Week 9 (PRE-BRONCHODILATOR) | | yyyy-mm-ddThh:mm | XX | XX |
| | Best FVC [L] | SCREENING (PRE-BRONCHODILATOR) | Y | yyyy-mm-ddThh:mm | xx | - |
| | | Week 5 (PRE-BRONCHODILATOR) | | yyyy-mm-ddThh:mm | XX | XX |
| | | Week 9 (PRE-BRONCHODILATOR) | | yyyy-mm-ddThh:mm | XX | XX |
| | FEV1 predicted [%] | SCREENING (PRE-BRONCHODILATOR) | Y | yyyy-mm-ddThh:mm | XX | - |
| | | Week 5 (PRE-BRONCHODILATOR) | | yyyy-mm-ddThh:mm | XX | XX |
| | | Week 9 (PRE-BRONCHODILATOR) | | yyyy-mm-ddThh:mm | XX | XX |
| | Best FEV1 [L] | SCREENING (POST-BRONCHODILATOR) | Y | yyyy-mm-ddThh:mm | XX | - |
| | | Week 5 (POST-BRONCHODILATOR) | | yyyy-mm-ddThh:mm | XX | XX |
| | | Week 9 (POST-BRONCHODILATOR) | | yyyy-mm-ddThh:mm | XX | XX |

>Sort order;

Subject Number, Parameter, Visit

- GTI 1401 11 Safety Analysis 11.7 Pregnancy Tests 11.7 Listing for Pregnancy Tests

| Subject | | Date of Sample | Date of Sample |
|---|---|---|---|
| Number | Visit | Collection | Test Result |
| xxxx | SCREENING<br>Week 5 | yyyy-mm-dd<br>yyyy-mm-dd | NEGATIVE<br>NEGATIVE |
| | Week 9 | yyyy-mm-dd | NEGATIVE |
| xxxx | SCREENING<br>Week 5<br>Week 9 | yyyy-mm-dd<br>yyyy-mm-dd<br>yyyy-mm-dd | NEGATIVE<br>NEGATIVE<br>NEGATIVE |

>Sort order; Subject Number, Visit

11 Safety Analysis

11.8 CT Scan

11.8 Listing for CT Scan

# Safety population

| Subject<br>Number | Visit | Date of Scan<br>Performed | Apparent Pulmonary<br>Emphysema Diagnosed | Was a CT Scan<br>performed | Lung Density [Unit] |
|---|---|---|---|---|---|
| XXXX | SCREENING | yyyy-mm-dd | Y | Y | XX.XX |
| XXXX | SCREENING | yyyy-mm-dd | N | Y | XX.XX |
| XXXX | SCREENING | yyyy-mm-dd | | N | XX.XX |

>Sort order;

Subject Number, Visit

>In this listing, if the record "not done" is exist in data, "not done" record will be presented.

- 11 Safety Analysis
  11.9 Physical Examination
  11.9 Listing for Physical Examination

# Safety population

| Subject | | | Category of Physical | Completion Status | |
|---|---|---|---|---|---|
| Number | Visit | Date of Examination | Examination | for Examination | Reason for Abnormal or Not Done |
| XXXX | SCREENING | yyyy-mm-dd | GENERAL | Y | _ |
| | | | APPEARANCE | | |
| | | | HEENT | Y | |
| | | | CARDIOVASCULAR | N | xxxxxxxxxxxxxxxxxxxxxxxx |
| | | | RESPIRATORY | Y | |
| | | | ABDOMINAL | Y | |
| | | | SKIN | Y | |
| | | | EXTREMITIES | Y | |
| | | | NEUROLOGIC | Y | |
| | | | MUSCULOSKELETAL | Y | |
| | | | LYMPHATIC | Y | |
| | | | OTHER / | | |
| | | | XXXXXXXXXXXXXX | Y | |
| | Week 9 | yyyy-mm-dd | GENERAL | | |
| | | | APPEARANCE | Y | |
| | | | HEENT | Y | |
| | | | CARDIOVASCULAR | Y | |
| | | | RESPIRATORY | Y | |
| | | | ABDOMINAL | Y | |
| | | | SKIN | Y | |
| | | | EXTREMITIES | Y | |
| | | | NEUROLOGIC | Y | |
| | | | MUSCULOSKELETAL | Y | |
| | | | LYMPHATIC | Y | |
| | | | OTHER / | | |
| | | | XXXXXXXXXXXXXXX | Y | |

- 11 Safety Analysis 11.9 Physical Examination
- 11.9 Listing for Physical Examination

Safety population

| Subject | | | Category of Physical | Completion Status | |
|---|---|---|---|---|---|
| Number | Visit | Date of Examination | Examination | for Examination | Reason for Abnormal or Not Done |

>Sort order;

Subject Number, Visit, Category of Physical Examination

>In this listing, if the record "not done" is exist in data, "not done" record will be presented.